CLINICAL TRIAL: NCT01648140
Title: A Phase II Multicenter, Parallel-Group, Randomized, Dose-Ranging Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Following 12 Weeks of Oral Administration of GSK2336805 With Pegylated Interferon and Ribavirin in Treatment-Naïve Subjects With Chronic Genotype 1 or 4 Hepatitis C Infection
Brief Title: Dose Ranging of GSK2336805 in Combination Therapy
Acronym: HAI115879
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115879
Record Dates: First submitted 2012-07-12; First posted 2012-07-24 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
Keywords: Genotype 4; GSK2336805; pegylated interferon; telaprevir; Genotype 1; chronic hepatitis C; ribavirin; NS5A inhibitor; hepatitis C virus (HCV) infection
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Infections | interventions — GSK2336805; peginterferon alfa-2a; Ribavirin; telaprevir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- T40 (Experimental): Hepatitis C virus (HCV) genotype 1 GSK2336805 40 mg, pegylated interferon alpha-2a, and ribavirin arm
  Interventions: Drug: GSK2336805 40 mg; Drug: Pegylated interferon alpha-2a; Drug: Ribavirin
- T60 (Experimental): Hepatitis C virus (HCV) genotype 1 GSK2336805 60 mg, pegylated interferon alpha-2a, and ribavirin arm
  Interventions: Drug: GSK2336805 60 mg; Drug: Pegylated interferon alpha-2a; Drug: Ribavirin
- PRT (Active Comparator): Hepatitis C virus (HCV) genotype 1 Telaprevir, pegylated interferon alpha-2a, and ribavirin arm
  Interventions: Drug: Pegylated interferon alpha-2a; Drug: Ribavirin; Drug: Telaprevir
- G4 (Experimental): Hepatitis C virus (HCV) genotype 4 GSK2336805 60 mg, pegylated interferon alpha-2a, and ribavirin arm
  Interventions: Drug: GSK2336805 60 mg; Drug: Pegylated interferon alpha-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: GSK2336805 40 mg — 20 mg tablet, round, 10-mm diameter, white to off-white, no markings
  Arms: T40
Drug: GSK2336805 60 mg — 30 mg tablet, round, 10-mm diameter, white to off-white, no markings
  Arms: G4; T60
Drug: Pegylated interferon alpha-2a — 180 microgram per 0.5 mL prefilled syringe for single use
  Other Names: Pegasys
Drug: Ribavirin — 200-mg tablet, capsule-shaped, light blue, film-coated, and debossed with "200" on 1 side and the logo "3RP" on the other side
  Other Names: Ribasphere
Drug: Telaprevir — 375 mg film-coated tablet
  Other Names: Incivek (United States); Incivo (European Union)
  Arms: PRT

SUMMARY:
GSK2336805 is a novel hepatitis C virus (HCV) non-structural 5A (NS5A) inhibitor being developed for the treatment of chronic HCV infection. This Phase II, multicenter, parallel-group, randomized, dose-ranging study will assess the safety and tolerability, antiviral activity, and pharmacokinetics of GSK2336805 at 2 dose levels (40 and 60 mg) in combination with pegylated interferon alfa-2a (PEG) and ribavirin (RIBA) in approximately 100 treatment-naïve subjects with chronic genotype 1 HCV infection.

In a separate nonrandomized single-arm cohort, up to 15 treatment-naïve subjects with genotype 4 chronic HCV infection will be enrolled in parallel at the dose level of 60 mg of GSK2336805.

DETAILED DESCRIPTION:
Subjects with chronic genotype 1 hepatitis C virus (HCV) infection will be randomly assigned on a 2:2:1 basis to 1 of 3 treatment arms: T40 (GSK2336805 40 mg and PEG + RIBA) or T60 (GSK2336805 60 mg and PEG + RIBA) or PEG + RIBA and telaprevir (PRT). Randomization will be stratified by interleukin 28B (IL28B) rs12979860 status (C/C versus carriage of the T allele), HCV genotype (1a vs. 1b), and plasma HCV Ribonucleic Acid (RNA) (<800,000 IU/mL versus ≥800,000 IU/mL).

An additional nonrandomized single-arm cohort of subjects with chronic genotype 4 HCV infection will be enrolled in parallel. A maximum of 15 genotype 4 subjects will receive GSK2336805 60 mg and PEG + RIBA. The purpose of this cohort is to further characterize the antiviral activity of GSK2336805 in subjects with chronic genotype 4 HCV infection. The schedule of assessments for the genotype 4 subjects will be the same as for the genotype 1 subjects. Recruitment of the genotype 4 subjects may be terminated when the target sample of genotype 1 subjects have been randomized.

Subjects in a GSK2336805 treatment arm who achieve extended rapid virologic response (eRVR) will receive a total of 24 weeks of therapy (12 weeks GSK2336805 in combination with PEG + RIBA followed by 12 weeks PEG + RIBA). Subjects who are HCV detectable at Week 4 and then undetectable at Week 12 will receive a total of 48 weeks of therapy (12 weeks GSK2336805 in combination with PEG + RIBA followed by 36 weeks PEG + RIBA). Subjects in the telaprevir treatment control arm will be managed according to the current product label for treatment-naïve subjects.

Subjects who complete treatment will undergo follow-up monitoring for 24 weeks after completion of therapy. At the end of the 24-week follow-up visit, subjects will have completed their participation in the study. The total duration of the study will be 48 weeks for subjects who achieve eRVR at Week 12 and up to 72 weeks for subjects who do not achieve eRVR at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Male or female aged 18 to 70 years of age, inclusive, at Screening.
* Genotype 1 or genotype 4 hepatitis C virus (HCV) infection as assessed by Versant HCV Genotype assay 2.0 (LiPA).
* Chronic HCV infection documented by at least 1 measurement of serum HCV RNA greater than or equal to 100,000 IU/mL measured during Screening by the COBAS High Pure/COBAS TaqMan HCV Test v2.0 and at least one of the following:
* A positive anti-HCV antibody, HCV RNA, or HCV genotype test at least 6 months prior to Baseline (Day 1) together with positive HCV RNA and anti-HCV antibody tests at the time of Screening; or
* A positive HCV RNA test and anti-HCV antibody test at the time of Screening together with either a liver biopsy consistent with chronic HCV infection (or a liver biopsy performed before enrollment with evidence of chronic hepatitis C disease, such as the presence of fibrosis).
* Naïve to all HCV antiviral treatment(s), including, but not limited to, immunomodulatory and nucleoside/nucleotide treatments for chronic HCV infection.
* Agree to interleukin 28B (IL28B) genotyping.
* A subject, who, in the opinion of the investigator, is an appropriate candidate for pegylated interferon alpha-2a (PEG)/ribavirin (RIBA)/protease inhibitor combination therapy for genotype 1 subjects and PEG/RIBA combination therapy for genotype 4 subjects.
* Body mass index >18 kg/m2 but not exceeding 36 kg/m2.
* A liver biopsy obtained within 3 years (36 calendar months) prior to the Day 1 visit, with a fibrosis classification of noncirrhotic as judged by a local pathologist (defined as Knodell less than or equal to 3, Metavir less than or equal to 2, Ishak less than or equal to 4, or Batts and Ludwig less than or equal to 2). Both incomplete and transition to cirrhosis (e.g., Metavir score 3) are considered as cirrhosis. If no recent (<36 months) liver biopsy is available, a study-qualifying biopsy must be performed prior to Baseline (Day 1).
* All fertile males and females must use 2 forms of effective contraception between them during treatment and during the 24 weeks after treatment ends.
* Females, is eligible to enter and participate in the study if of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) and includes any female who has had a hysterectomy or has had a bilateral oophorectomy (ovariectomy) or has had a bilateral tubal ligation or is postmenopausal (demonstrate total cessation of menses for greater than 1 year).
* Females, is eligible to enter and participate in the study if of childbearing potential and has a negative urine or serum pregnancy test at Screening and within the 24-hour period prior to the first dose of study medication and completely abstains from intercourse for 2 weeks before exposure to the study medication, throughout the clinical study, and for 24 weeks after completion or premature discontinuation from this study or uses 2 of the following acceptable methods of contraception throughout the clinical study and for 24 weeks after completion or premature discontinuation from this study:
* Any intrauterine device with a documented failure rate of <1% per year
* Double-barrier contraception (condom, diaphragm, or cervical cap used with spermicidal jelly)
* Male partner who is sterile prior to the female subject's study entry and is the sole sexual partner for that female
* Any other contraceptive method with a documented failure rate of <1% per year
* Otherwise healthy as determined by the medical history, physical examination, ECG findings, and clinical laboratory measurements performed at Screening.

Exclusion Criteria:

* Positive test at Screening visit for hepatitis B surface antigen (HBsAg) or antihuman immunodeficiency virus antibody
* History of any other clinically significant chronic liver disease (e.g., hemochromatosis, autoimmune hepatitis, Wilson's disease, 1-antitrypsin deficiency, alcoholic liver disease, >Grade 1 nonalcoholic steatohepatitis, and toxin exposures). Subjects with Gilbert's syndrome who otherwise meet all inclusion/exclusion criteria are eligible.
* History of ascites, variceal hemorrhage, hepatic encephalopathy, or conditions consistent with decompensated liver disease
* Positive results on urine screen for drugs of abuse test at Screening (unless used as medical treatment, e.g., with a prescription)
* History of alcohol/drug abuse or dependence within 6 months of the study start (unless participating in a controlled rehabilitation program)
* Screening visit electrocardiogram corrected QT (QTc) interval value >450 ms and/or clinically significant electrocardiogram findings
* Personal or family history of Torsade de Pointes findings
* Pregnant or nursing
* Male with a female partner who is pregnant
* Abnormal hematological and biochemical parameters, including:
* Neutrophil count <1500 cells/mm3 (or <1250 cells/mm3 for African American/Black subjects)
* Hemoglobin <11 g/dL in females or <12 g/dL in males
* Creatinine greater than or equal to 1.5 × the upper limit of normal (ULN)
* Estimated creatinine clearance less than or equal to 50 mL/min (as calculated using the Cockcroft-Gault formula)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase greater than or equal to 5 × ULN
* Total bilirubin greater than or equal to 2.0 × ULN (except subjects with Gilbert's syndrome)
* Albumin less than or equal to 3.0 g/dL
* Platelet count less than or equal to 90,000/mm3
* History of major organ transplantation with an existing functional graft
* Thyroid dysfunction not adequately controlled
* History of suicide attempt or hospitalization for depression in the past 5 years
* History of any current (within 6 months) severe or poorly controlled psychiatric disorder
* Subjects who have had a severe or poorly controlled psychiatric disorder more than 6 months ago but less than 5 years ago are eligible for study participation but must be assessed and followed (if recommended) by a mental health professional.
* History or current evidence of immunologic disorder; cardiac or pulmonary disease; seizure disorder; or cancer or history of malignancy that in the opinion of the investigator makes the subject unsuitable for the study.
* Treated with herbal or natural remedies with antiviral activity within 30 days of the baseline visit or has a history of having received any systemic antineoplastic or immunomodulatory treatment (including mycophenolate mofetil, thymosin alpha, supraphysiologic doses of steroids >10 mg/day and radiation) within 6 months of the baseline visit or expects that such treatment will be needed at any time during the study.
* Participated in a clinical study with an investigational drug, biologic, or device within 3 months prior to the first dose administration.
* History of a known allergy to antiviral medications, including telaprevir, pegylated interferon alpha-2a (PEG), ribavirin (RIBA), or any excipient in the investigational product or history of drug or other allergy that, in the opinion of the investigator, contradicts participation.
* Requires prohibited medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2012-08-01; Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (32):
- United States (18):
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Brockton, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Jenkintown, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Annandale, Virginia
  - GSK Investigational Site, Norfolk, Virginia
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Liège
- Bulgaria (2):
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- France (3):
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
- Germany (5):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Puerto Rico (2):
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Protocol contains no citations
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 115879 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115879 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115879 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115879 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115879 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115879 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across 29 centers in 6 countries (United States, Puerto Rico, Germany, Belgium, France, and Bulgaria) from 15 August 2012 to 16 July 2014.
Pre-assignment Details: Participants with treatment-naïve(TN) chronic genotype1(G1) hepatitis C virus (HCV) infection were randomly allocated on 2:2:1 basis to 2 dose levels of GSK2336805 or telaprevir. In a nonrandomized single-arm cohort, participants with TN genotype4(G4) chronic HCV infection were enrolled in parallel at dose level of 60 milligrams (mg) of GSK2336805.
Groups:
- GSK2336805 40 mg, G1 HCV: Participants with chronic G1 HCV infection received GSK2336805 40 mg orally (20 mg x 2 tablets) once daily in the morning with food in combination with antiviral therapy (Pegylated Interferon Alfa-2a [PEG] + Ribavirin [RIBA]) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on the extended rapid virologic response (eRVR) achievement. PEG dose was 180 micrograms (µg) once weekly subcutaneous (SC) injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kilogram [kg]) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken in 2 divided doses with food.
- GSK2336805 60 mg, G1 HCV: Participants with chronic G1 HCV infection received GSK2336805 60 mg orally (30 mg x 2 tablets) once daily in the morning with food in combination with antiviral therapy (PEG+RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was 180 µg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken orally in 2 divided doses with food.
- Telaprevir, G1 HCV: Participants with chronic G1 HCV infection received two telaprevir 375 mg tablets orally 3 times a day (7 to 9 hours apart) with food containing approximately 20 grams of fat in combination with antiviral therapy (PEG+RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was 180 µg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken orally in 2 divided doses with food.
- GSK2336805 60 mg, G4 HCV: Participants with chronic G4 HCV infection received GSK2336805 60 mg orally (30 mg x 2 tablets) once daily in the morning with food in combination with antiviral therapy (PEG+RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was 180 µg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken orally in 2 divided doses with food.
Period: Overall Study
Arm/Group | GSK2336805 40 mg, G1 HCV | GSK2336805 60 mg, G1 HCV | Telaprevir, G1 HCV | GSK2336805 60 mg, G4 HCV
Started | 41 | 40 | 17 | 13
Completed | 29 | 28 | 9 | 11
Not Completed | 12 | 12 | 8 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 7 | 1 | 0
Not completed — Adverse Event | 3 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 3 | 2
Not completed — Lost to Follow-up | 2 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK2336805 40 mg, Genotype 1 HCV: Participants with chronic G1 HCV infection received GSK2336805 40 mg orally (20 mg x 2 tablets) once daily in the morning with food in combination with antiviral therapy (PEG + RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on the eRVR achievement. PEG dose was 180 µg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken in 2 divided doses with food.
- GSK2336805 60 mg, Genotype 1 HCV: Participants with chronic G1 HCV infection received GSK2336805 60 mg orally (30 mg x 2 tablets) once daily in the morning with food in combination with antiviral therapy (PEG+RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was 180 µg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken orally in 2 divided doses with food.
- Telaprevir, Genotype 1 HCV: Participants with chronic G1 HCV infection received two telaprevir 375 mg tablets orally 3 times a day (7 to 9 hours apart) with food containing approximately 20 grams of fat in combination with antiviral therapy (PEG+RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was 180 µg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken orally in 2 divided doses with food.
- GSK2336805 60 mg, Genotype 4 HCV: Participants with chronic G4 HCV infection received GSK2336805 60 mg orally (30 mg x 2 tablets) once daily in the morning with food in combination with antiviral therapy (PEG+RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was 180 µg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken orally in 2 divided doses with food.
- Total: Total of all reporting groups
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV | Total
Number analyzed (Participants) | 41 | 40 | 17 | 13 | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (13.23) | 40.8 (9.87) | 39.4 (12.02) | 45.3 (11.46) | 42.2 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 6 | 3 | 38
  Male | 28 | 24 | 11 | 10 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 2 | 3 | 17
  White | 34 | 33 | 15 | 9 | 91
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving eRVR
Description: eRVR is defined as plasma HCV ribonucleic acid (RNA) <lower limit of quantification (LLOQ) and target not detected at Weeks 4 and 12. Participants who discontinued prior to Week 12 assessments or had missing HCV RNA values at Weeks 4 and 12 were treated as non-responders.
Time Frame: Week 4 and Week 12
Population: Intent-To-Treat (ITT) Population: comprised of all participants who met the study criteria and were randomly assigned to treatment in the study with documented evidence of having received at least 1 dose of randomized treatment and at least 1 post Baseline HCV RNA measurement.
Measure: Number; unit: Participants
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Participants | 23 | 21 | 9 | 9

2. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Any Serious Adverse Events (SAEs) up to Week 12
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign(including an abnormal laboratory finding), symptom, or disease(new or exacerbated) temporally associated with the use of a medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, a congenital anomaly/birth defect, important medical events that jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition.
Time Frame: From the start of study treatment up to Week 12
Population: Safety Population: comprised of all participants who received at least 1 dose of study medication (GSK2336805 or telaprevir).
Measure: Number; unit: Participants
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Participants
  Any AE | 39 | 37 | 17 | 13
  Any SAE | 0 | 2 | 3 | 1

3. Primary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Indicated Time Points up to Week 12
Description: Blood pressure measurements were taken to observe vital signs and included SBP and DBP at the Baseline, Day 2, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and Post-treatment (PT) Follow Up (FU) Weeks 4, 12 and 24. Change from Baseline in SBP and DBP is summarized for each post-Baseline assessment up to Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) up to 12-week treatment period
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X,X,X,X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the safety population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Millimeters of mercury (mmHg)
  DBP; Day2; n=41, 40, 17, 13 | -1.2 (6.63) | -1 (7.03) | -3 (9.03) | -1.5 (10.45)
  DBP; Week1; n=41, 39, 15, 13 | -0.4 (7.98) | -2.2 (9.13) | 1 (10.54) | -1 (7.99)
  DBP; Week2; n=41, 39, 14, 13 | -0.4 (10.41) | -1.7 (9.52) | -0.3 (8.8) | -2.8 (11.09)
  DBP; Week4; n=41, 39, 14, 13 | -1.2 (7.73) | -4.4 (9.78) | -3.9 (9.74) | 0.8 (9.92)
  DBP; Week6; n=41, 39, 13, 13 | -1.2 (7.65) | -4.8 (9.86) | -5.9 (7.82) | -1.6 (10.1)
  DBP; Week8; n=41, 39, 13, 13 | -2.1 (10) | -2.9 (9.11) | -4.4 (7.63) | -2.4 (9.02)
  DBP; Week12; n=38, 35, 12, 13 | 0.3 (8.48) | -4.4 (10.24) | -3.5 (9.2) | -1 (9.11)
  SBP; Day2; n=41, 40, 17, 13 | -1.4 (10.1) | -0.8 (12.85) | -3.3 (10.46) | -1.3 (13.95)
  SBP; Week1; n=41, 39, 15, 13 | 0.9 (12.99) | -3 (11.24) | -4.5 (12.67) | -2.6 (11.84)
  SBP; Week2; n=41, 39, 14, 13 | -2 (10.57) | -0.7 (11.67) | -4.1 (12.67) | -4.2 (17.35)
  SBP; Week4; n=41, 39, 14, 13 | -3.6 (11.56) | -4.2 (16.2) | -3.8 (9.73) | -5.2 (15.3)
  SBP; Week6; n=41, 39, 13, 13 | -0.4 (14.47) | -3.8 (13.28) | -5.9 (11.39) | 0.2 (14.47)
  SBP; Week8; n=41, 39, 13, 13 | -3.7 (12.15) | -1.5 (12.64) | -2.9 (10.36) | -4.2 (12.95)
  SBP; Week12; n=38, 35, 12, 13 | -1.9 (13.65) | -1.4 (11.72) | -5.2 (5.81) | -2.6 (19.16)

4. Primary Outcome: Mean Change From Baseline in Heart Rate at the Indicated Time Points up to Week 12
Description: Vital sign monitoring included heart rate, measured at the Baseline, Day 2, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4, 12 and 24. Change from Baseline in heart rate is summarized for each post-Baseline assessment upto Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Day 2, Weeks 1, 2, 4, 6, 8, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Beats per minute
  Heart Rate; Day2; n=41, 40, 17, 13 | 6.5 (8.65) | 5.4 (9.96) | 9.3 (11.74) | 3.8 (5.79)
  Heart Rate; Week1; n=41, 39, 15, 13 | 1.5 (8.33) | 3.1 (8.75) | 8.1 (6.32) | 7.7 (10.11)
  Heart Rate; Week2; n=41, 39, 14, 13 | 3.8 (9.02) | 4.2 (12.14) | 8.7 (8.17) | 7.8 (8.6)
  Heart Rate; Week4; n=41, 39, 14, 13 | 6.8 (9.42) | 4.2 (11.78) | 10.7 (11.39) | 5.5 (8.35)
  Heart Rate; Week6; n=41, 39, 13, 13 | 8 (10.15) | 5 (10.98) | 13.8 (9.75) | 10.2 (8.2)
  Heart Rate; Week8; n=41, 39, 13, 13 | 4.7 (9.91) | 6.8 (12.42) | 14.2 (10.36) | 12.8 (12.27)
  Heart Rate; Week12; n=38, 35, 12, 13 | 7 (9.2) | 5.3 (12.1) | 11 (8.02) | 8.4 (9.47)

5. Primary Outcome: Mean Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count and White Blood Cell Count at the Indicated Time Points up to Week 12
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelet count and white blood cell count at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4. Change from Baseline in the basophils, eosinophils, lymphocytes, total neutrophils, platelet count and white blood cell count values are summarized for each post-Baseline assessment until Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6, 8 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Giga cells per liter
  Basophils; Week1; n=38, 38, 14, 11 | -0.011 (0.0191) | -0.011 (0.0193) | -0.012 (0.0105) | -0.013 (0.0119)
  Basophils; Week2; n=40, 38, 14, 10 | -0.014 (0.0175) | -0.01 (0.0192) | -0.009 (0.0107) | -0.009 (0.0179)
  Basophils; Week4; n=41, 38, 14, 13 | -0.017 (0.0184) | -0.012 (0.0187) | -0.01 (0.0118) | -0.015 (0.0113)
  Basophils; Week6; n=41, 37, 12, 12 | -0.015 (0.021) | -0.013 (0.0205) | -0.013 (0.0114) | -0.013 (0.0106)
  Basophils; Week8; n=38, 39, 13, 13 | -0.019 (0.0155) | -0.016 (0.018) | -0.009 (0.0132) | -0.012 (0.0142)
  Basophils; Week12; n=37, 36, 12, 12 | -0.018 (0.0184) | -0.013 (0.0187) | -0.011 (0.0124) | -0.012 (0.0153)
  Eosinophils; Week1; n=38, 38, 14, 11 | -0.051 (0.0874) | -0.075 (0.106) | -0.059 (0.0578) | -0.085 (0.1052)
  Eosinophils; Week2; n=40, 38, 14, 10 | -0.08 (0.1004) | -0.111 (0.0912) | -0.059 (0.104) | -0.114 (0.1247)
  Eosinophils; Week4; n=41, 38, 14, 13 | -0.105 (0.0872) | -0.132 (0.1057) | -0.079 (0.1089) | -0.108 (0.0923)
  Eosinophils; Week6; n=41, 37, 12, 12 | -0.117 (0.0929) | -0.134 (0.1182) | -0.113 (0.0607) | -0.109 (0.1208)
  Eosinophils; Week8; n=38, 39, 13, 13 | -0.121 (0.0897) | -0.134 (0.1061) | -0.13 (0.0965) | -0.104 (0.0916)
  Eosinophils; Week12; n=37, 36, 12, 12 | -0.118 (0.0916) | -0.112 (0.1594) | -0.106 (0.1152) | -0.102 (0.1428)
  Lymphocytes; Week1; n=38, 38, 14, 11 | -0.319 (0.5006) | -0.282 (0.5698) | -0.608 (0.5466) | -0.371 (0.4332)
  Lymphocytes; Week2; n=40, 38, 14, 10 | -0.448 (0.5385) | -0.603 (0.5921) | -0.675 (0.5639) | -0.553 (0.4346)
  Lymphocytes; Week4; n=41, 38, 14, 13 | -0.787 (0.5055) | -0.854 (0.5114) | -0.989 (0.5293) | -0.773 (0.4104)
  Lymphocytes; Week6; n=41, 37, 12, 12 | -0.963 (0.5313) | -1.043 (0.5928) | -1.334 (0.4906) | -0.93 (0.4955)
  Lymphocytes; Week8; n=38, 39, 13, 13 | -0.953 (0.4624) | -1.061 (0.6021) | -1.256 (0.3509) | -0.964 (0.5098)
  Lymphocytes; Week12; n=37, 36, 12, 12 | -1.118 (0.5139) | -1.074 (0.5883) | -1.438 (0.4773) | -1.048 (0.6612)
  Monocytes; Week1; n=38, 38, 14, 11 | -0.103 (0.1418) | -0.056 (0.145) | 0.034 (0.1502) | -0.025 (0.0808)
  Monocytes; Week2; n=40, 38, 14, 10 | -0.122 (0.227) | -0.061 (0.1785) | -0.091 (0.1562) | -0.034 (0.1687)
  Monocytes; Week4; n=41, 38, 14, 13 | -0.151 (0.1771) | -0.129 (0.158) | -0.126 (0.1471) | -0.055 (0.2103)
  Monocytes; Week6; n=41, 37, 12, 12 | -0.182 (0.1664) | -0.171 (0.1326) | -0.245 (0.1786) | -0.135 (0.1088)
  Monocytes; Week8; n=38, 39, 13, 13 | -0.229 (0.167) | -0.165 (0.1779) | -0.185 (0.1344) | -0.124 (0.2164)
  Monocytes; Week12; n=37, 36, 12, 12 | -0.185 (0.1715) | -0.183 (0.1438) | -0.219 (0.1493) | -0.133 (0.2048)
  Total Neutrophils; Week1; n=38, 38, 14, 11 | -2.338 (1.4959) | -1.871 (1.5089) | -1.158 (1.2688) | -1.378 (0.598)
  Total Neutrophils; Week 2; n=40, 38, 14, 10 | -2.114 (1.9189) | -2.121 (1.6445) | -1.186 (1.3343) | -1.468 (0.584)
  Total Neutrophils; Week4; n=41, 38, 14, 13 | -2.487 (1.9145) | -2.333 (1.5497) | -1.412 (1.5704) | -1.603 (0.5953)
  Total Neutrophils; Week6; n=41, 37, 12, 12 | -2.51 (1.8144) | -2.247 (1.5132) | -1.413 (1.4303) | -1.683 (0.661)
  Total Neutrophils; Week8; n=38, 39, 13, 13 | -2.706 (1.7553) | -2.168 (1.6902) | -1.222 (1.3481) | -1.613 (0.6882)
  Total Neutrophils; Week12; n=37, 36, 12, 12 | -2.894 (1.8124) | -2.188 (1.7297) | -1.649 (0.8749) | -1.483 (0.5873)
  Platelet Count; Week1; n=38, 39, 14, 11 | -58.5 (36.23) | -51.4 (36.42) | -59.5 (36.29) | -33.1 (33.32)
  Platelet Count; Week2; n=41, 38, 14, 11 | -58 (43.92) | -57.8 (44.02) | -41.4 (37.44) | -34.4 (41.74)
  Platelet Count; Week4; n=41, 38, 14, 13 | -54.4 (49.18) | -55.9 (47.19) | -56.2 (50.99) | -33.8 (61.79)
  Platelet Count; Week6; n=41, 38, 12, 13 | -66.8 (50.43) | -71.9 (38.6) | -71.3 (47.07) | -46 (46.05)
  Platelet Count; Week8; n=39, 39, 13, 13 | -74.9 (42.31) | -75.7 (45.82) | -60.1 (43.26) | -52.6 (43.54)
  Platelet Count; Week12; n=38, 34, 12, 12 | -73.4 (45.3) | -85.3 (40.42) | -58.8 (58.77) | -53 (39.49)
  White Blood Cell count; Week1; n=38, 38, 14, 11 | -2.83 (1.705) | -2.3 (1.872) | -1.81 (1.516) | -1.87 (0.508)
  White Blood Cell count; Week2; n=40, 38, 14, 10 | -2.77 (2.178) | -2.92 (1.81) | -2.01 (1.869) | -2.17 (0.886)
  White Blood Cell count; Week4; n=41, 38, 14, 13 | -3.55 (2.183) | -3.47 (1.712) | -2.61 (2.055) | -2.55 (0.919)
  White Blood Cell count; Week6; n=41, 37, 12, 12 | -3.78 (2.051) | -3.62 (1.682) | -3.09 (1.69) | -2.85 (0.923)
  White Blood Cell count; Week8; n=38, 39, 13, 13 | -4.03 (2.028) | -3.55 (1.896) | -2.8 (1.477) | -2.8 (1.04)
  White Blood Cell count; Week12; n=37, 36, 12, 12 | -4.33 (2.149) | -3.58 (1.934) | -3.42 (1.104) | -2.77 (0.963)

6. Primary Outcome: Mean Change From Baseline in Red Blood Cell Count at the Indicated Time Points up to Week 12
Description: Blood samples were collected for the measurement of red blood cell count at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4. Change from Baseline in the red blood cell count values are summarized for each post-Baseline assessment until Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6, 8 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Trillion cells per liter
  Red Blood Cell count; Week1; n=38, 39, 14, 12 | -0.15 (0.226) | -0.04 (0.279) | -0.18 (0.212) | -0.13 (0.303)
  Red Blood Cell count; Week2; n=41, 38, 14, 12 | -0.48 (0.376) | -0.44 (0.508) | -0.57 (0.312) | -0.28 (0.361)
  Red Blood Cell count; Week4; n=41, 38, 14, 13 | -0.88 (0.507) | -0.64 (0.623) | -1.03 (0.441) | -0.72 (0.559)
  Red Blood Cell count; Week6; n=41, 38, 12, 13 | -0.97 (0.504) | -0.78 (0.563) | -1.28 (0.49) | -0.86 (0.52)
  Red Blood Cell count; Week8; n=39, 39, 13, 13 | -1.01 (0.506) | -0.82 (0.534) | -1.45 (0.357) | -0.85 (0.412)
  Red Blood Cell count; Week12; n=38, 36, 12, 12 | -1.08 (0.48) | -0.79 (0.56) | -1.61 (0.464) | -0.92 (0.459)

7. Primary Outcome: Mean Change From Baseline in Hemoglobin at the Indicated Time Points up to Week 12
Description: Blood samples were collected for the measurement of hemoglobin at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Week 4. Change from Baseline in the hemoglobin values are summarized for each post-Baseline assessment until Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6, 8 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Grams per liter
  Hemoglobin; Week1; n=38, 39, 14, 12 | -5.2 (6.98) | -2.3 (9.38) | -6.6 (5.83) | -5.3 (8.85)
  Hemoglobin; Week2; n=41, 38, 14, 12 | -16.7 (12.54) | -14.9 (16.21) | -20.5 (10.66) | -9.9 (11.5)
  Hemoglobin; Week4; n=41, 38, 14, 13 | -28.6 (15.38) | -22.1 (18.98) | -34.4 (13.55) | -22.5 (14.89)
  Hemoglobin; Week6; n=41, 38, 12, 13 | -30.1 (14.54) | -24.7 (16) | -40.8 (14.11) | -25.2 (12.28)
  Hemoglobin; Week8; n=39, 39, 13, 13 | -30.5 (13.29) | -25.5 (14.22) | -44.9 (11.73) | -25.2 (8.66)
  Hemoglobin; Week12; n=38, 36, 12, 12 | -33 (12.88) | -24.1 (13.41) | -47.4 (14.12) | -27.6 (12.05)

8. Primary Outcome: Mean Change From Baseline in Hematocrit at the Indicated Time Points up to Week 12
Description: Blood samples were collected for the measurement of hematocrit at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Week 4. Change from Baseline in the hematocrit values are summarized for each post-Baseline assessment until Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6, 8 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Ratio
  Hematocrit; Week1; n=38, 39, 14, 12 | -0.0196 (0.02345) | -0.0069 (0.02751) | -0.0201 (0.01921) | -0.0166 (0.0298)
  Hematocrit; Week2; n=41, 38, 14, 12 | -0.0539 (0.03653) | -0.0465 (0.04738) | -0.0609 (0.03007) | -0.0335 (0.03625)
  Hematocrit; Week4; n=41, 38, 14, 13 | -0.0848 (0.04576) | -0.0621 (0.05468) | -0.0999 (0.03967) | -0.0668 (0.04445)
  Hematocrit; Week6; n=41, 38, 12, 13 | -0.0859 (0.0411) | -0.0685 (0.04487) | -0.1203 (0.04463) | -0.074 (0.03316)
  Hematocrit; Week8; n=39, 39, 13, 13 | -0.0838 (0.03955) | -0.0663 (0.04144) | -0.1235 (0.03288) | -0.07 (0.02758)
  Hematocrit; Week12; n=38, 36, 12, 12 | -0.0843 (0.04038) | -0.0589 (0.03648) | -0.1318 (0.03847) | -0.0688 (0.03298)

9. Primary Outcome: Mean Change From Baseline in Mean Corpuscle Volume at the Indicated Time Points up to Week 12
Description: Blood samples were collected for the measurement of mean corpuscle volume at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4. Change from Baseline in the mean corpuscle volume values are summarized for each post-Baseline assessment until Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6, 8 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Femtoliters
Groups:
- GSK2336805 60 mg, Genotype 1 HCV: Participants with chronic G1 HCV infection received GSK2336805 60 mg orally (30 mg x 2 tablets) OD in the morning with food in combination with antiviral therapy (PEG+RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was 180 µg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken orally in 2 divided doses with food.
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Femtoliters
  Mean corpuscle volume; Week1; n=38, 39, 14, 12 | -1.1 (1.21) | -0.8 (1.37) | -0.4 (1.15) | -0.7 (1.37)
  Mean corpuscle volume; Week2; n=41, 38, 14, 12 | -2 (1.84) | -1.4 (1.59) | -1.4 (1.09) | -1.5 (1.45)
  Mean corpuscle volume; Week4; n=41, 38, 14, 13 | 0.3 (3.33) | 0.2 (3.4) | -0.8 (1.58) | -0.2 (2.94)
  Mean corpuscle volume; Week6; n=41, 38, 12, 13 | 2.3 (4.76) | 1.8 (4.67) | -0.2 (2.37) | 1.4 (4.63)
  Mean corpuscle volume; Week8; n=39, 39, 13, 13 | 3.8 (5.39) | 3 (5.2) | 3.1 (2.78) | 2.2 (3.75)
  Mean corpuscle volume; Week12; n=38, 34, 12, 12 | 5.7 (6) | 4.2 (6.3) | 5.3 (4.14) | 3.8 (4.28)

10. Primary Outcome: Mean Change From Baseline in Albumin at the Indicated Time Points up to Week 12
Description: Blood samples were collected for the measurement of albumin at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4. Change from Baseline in the albumin values are summarized for each post-Baseline assessment until Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6, 8 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Grams per liter
  Albumin; Week1; n=40, 39, 15, 13 | -0.6 (2.67) | -0.3 (2.46) | -1.1 (1.6) | -1 (1.87)
  Albumin; Week2; n=41, 38, 14, 13 | -1.3 (2.98) | -1.5 (2.68) | -2 (2.6) | -0.2 (2.39)
  Albumin; Week4; n=41, 39, 14, 13 | -1.9 (2.48) | -1.5 (2.52) | -3 (3.21) | -1.2 (1.46)
  Albumin; Week6; n=41, 38, 13, 13 | -2.2 (2.65) | -1.5 (2.27) | -3.5 (3.36) | -2.1 (2.22)
  Albumin; Week8; n=40, 39, 13, 13 | -2.6 (2.99) | -1.7 (2) | -3.7 (4.71) | -1.5 (1.94)
  Albumin; Week12; n=37, 35, 12, 13 | -2.1 (3.03) | -1.3 (2.84) | -3.3 (3.02) | -1.6 (2.1)

11. Primary Outcome: Mean Change From Baseline in Alkaline Phosphatase (ALP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Creatine Kinase (CK) and Gamma Glutamyl Transferase (GGT) at the Indicated Time Points up to Week 12
Description: Blood samples were collected for the measurement of ALP, ALT, AST, CK and GGT at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4 Change from Baseline in the ALP, ALT, AST, CK and GGT values are summarized for each post-Baseline assessment until Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6, 8 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
International units per liter
  ALP; Week1; n=40, 39, 15, 13 | 0 (7.73) | 1.5 (10.21) | 3.9 (19.36) | -0.2 (17.45)
  ALP; Week2; n=41, 38, 14, 13 | 4.6 (9.26) | 3.8 (16.22) | 9.4 (21.15) | 3.8 (12.43)
  ALP; Week4; n=41, 39, 14, 13 | 8.6 (11.12) | 7.1 (13.76) | 11.7 (26.61) | 7.2 (15.3)
  ALP; Week6; n=41, 38, 13, 13 | 9.1 (13.73) | 7.2 (17.1) | 16.6 (31.03) | 6.6 (16.38)
  ALP; Week8; n=40, 39, 13, 13 | 6.9 (15.59) | 6.5 (15.91) | 15.5 (25.83) | 5.6 (14.72)
  ALP; Week12; n=37, 35, 12, 13 | 6.7 (15.56) | 6.4 (20.78) | 11.7 (25.09) | 7.3 (18.33)
  ALT; Week1; n=40, 39, 15, 13 | -26.8 (31.64) | -24.4 (32.39) | -30.7 (30.1) | -25.6 (20.74)
  ALT; Week2; n=41, 38, 14, 13 | -28.2 (40.33) | -24.9 (47.49) | -35.4 (36.38) | -26.8 (24.25)
  ALT; Week4; n=41, 39, 14, 13 | -32.5 (44.5) | -25.3 (50.87) | -40.4 (38.73) | -33 (28.79)
  ALT; Week6; n=41, 38, 13, 13 | -36 (49.77) | -30.3 (50.74) | -40.8 (41.51) | -38.4 (29.11)
  ALT; Week8; n=40, 39, 13, 13 | -36.8 (55.75) | -25.4 (55.92) | -39.9 (40.27) | -39.5 (29.92)
  ALT; Week12; n=37, 35, 12, 13 | -38.9 (59.7) | -23.5 (59.69) | -43.7 (40.45) | -36.8 (24.75)
  AST; Week1; n=40, 39, 15, 13 | -12.3 (16.28) | -15.2 (21.55) | -18.1 (21.77) | -13.9 (10.52)
  AST; Week2; n=41, 38, 14, 13 | -10 (20.84) | -11.6 (26.3) | -18.4 (23.52) | -10.2 (12.56)
  AST; Week4; n=41, 39, 14, 13 | -12.8 (21.45) | -10.6 (27.4) | -20.9 (25.86) | -15.8 (11.92)
  AST; Week6; n=41, 38, 13, 13 | -13.8 (21.56) | -13.8 (25.01) | -21.6 (28.43) | -19.5 (12.99)
  AST; Week8; n=40, 39, 13, 13 | -13.1 (26.01) | -7.6 (38.38) | -21.8 (26.38) | -18.6 (12.38)
  AST; Week12; n=37, 35, 12, 13 | -14.4 (25.58) | -6.5 (36.17) | -25.7 (27.32) | -17.3 (12.68)
  CK; Week1; n=40, 39, 15, 13 | 18.2 (82.13) | -10.9 (103.31) | -3.3 (32.1) | -43.5 (82.73)
  CK; Week2; n=41, 38, 14, 13 | -0.7 (53.87) | -22.6 (77.26) | -9.6 (36.26) | -28.5 (54.43)
  CK; Week4; n=41, 39, 14, 13 | 4.5 (141.46) | -32.1 (59.61) | -14.4 (22.06) | -47.7 (59.52)
  CK; Week6; n=41, 38, 13, 13 | -26 (63.11) | 56.1 (566.79) | -21.5 (48.49) | -64.5 (110.82)
  CK; Week8; n=40, 39, 13, 13 | -21.3 (95.03) | -33.2 (65.96) | -30.3 (51.17) | -66.8 (107.3)
  CK; Week12; n=37, 35, 12, 13 | -36.3 (75.56) | -33.9 (47.72) | -20.9 (59.82) | -48.5 (61.63)
  GGT; Week1; n=40, 39, 15, 13 | -3.7 (20.79) | -2 (16.83) | -10.3 (19.38) | -6.4 (23.77)
  GGT; Week2; n=41, 38, 14, 13 | -11.7 (33.78) | -17.1 (45.23) | -19.9 (29.59) | -7.2 (29.11)
  GGT; Week4; n=41, 39, 14, 13 | -24.5 (52.93) | -25.5 (59.64) | -27.7 (36.64) | -16.2 (36.59)
  GGT; Week6; n=41, 38, 13, 13 | -28.1 (67.33) | -30.5 (72.27) | -30.5 (44.3) | -23.8 (39.91)
  GGT; Week8; n=40, 39, 13, 13 | -32.1 (70.41) | -27.2 (80.33) | -30.5 (45.05) | -28.5 (45.5)
  GGT; Week12; n=37, 35, 12, 13 | -29.7 (80.2) | -20.7 (73.43) | -33.6 (49.61) | -30 (53.44)

12. Primary Outcome: Mean Change From Baseline in Direct Bilirubin, Total Bilirubin and Creatinine at the Indicated Time Points up to Week 12
Description: Blood samples were collected for the measurement of direct bilirubin, total bilirubin and creatinine at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4. Change from Baseline in the direct bilirubin, total bilirubin and creatinine values are summarized for each post-Baseline assessment until Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6, 8 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Micromoles per liter
  Total Bilirubin; Week1; n=40, 39, 15, 13 | 6.9 (8.74) | 6.7 (8.93) | 8.1 (11.81) | 4.2 (8.36)
  Total Bilirubin; Week2; n=41, 38, 14, 13 | 5.8 (6.62) | 5.5 (6.84) | 5.6 (9.8) | 6.5 (9.34)
  Total Bilirubin; Week4; n=41, 39, 14, 13 | 2.2 (5.03) | 2.9 (3.52) | 0.7 (8.94) | 2.5 (5.97)
  Total Bilirubin; Week6; n=41, 38, 13, 13 | 1.5 (4.14) | 2.7 (3.97) | -0.5 (9.09) | 2.1 (6.87)
  Total Bilirubin; Week8; n=40, 39, 13, 13 | 1.4 (4.63) | 2.3 (4.93) | -0.3 (9.83) | 1.8 (6.39)
  Total Bilirubin; Week12; n=37, 35, 12, 13 | 0.4 (4.46) | 1.4 (5.61) | -2.8 (10.04) | 1.2 (5.31)
  Direct Bilirubin; Week1; n=1, 1, 1, 1 | 0 (NA) — A value of NA indicates not applicable | 2 (NA) — too few participants or number of participants were analyzed at the indicated test/time point. | -8 (NA) — too few participants or number of participants were analyzed at the indicated test/time point. | -1 (NA) — too few participants or number of participants were analyzed at the indicated test/time point.
  Direct Bilirubin; Week2; n=1, 1, 1, 1 | 0 (NA) — too few participants or number of participants were analyzed at the indicated test/time point. | 0 (NA) — too few participants or number of participants were analyzed at the indicated test/time point. | -14 (NA) — too few participants or number of participants were analyzed at the indicated test/time point. | 1 (NA) — too few participants or number of participants were analyzed at the indicated test/time point.
  Direct Bilirubin; Week4; n=1, 1, 0, 0 | 0 (NA) — too few participants or number of participants were analyzed at the indicated test/time point. | 2 (NA) — too few participants or number of participants were analyzed at the indicated test/time point. | NA (NA) — too few participants or number of participants were analyzed at the indicated test/time point. | NA (NA) — too few participants or number of participants were analyzed at the indicated test/time point.
  Direct Bilirubin; Week6; n=1, 1, 0, 0 | 0 (NA) — too few participants or number of participants were analyzed at the indicated test/time point. | 0 (NA) — too few participants or number of participants were analyzed at the indicated test/time point. | NA (NA) — too few participants or number of participants were analyzed at the indicated test/time point. | NA (NA) — too few participants or number of participants were analyzed at the indicated test/time point.
  Creatinine; Week1; n=40, 39, 15, 13 | -1.41 (5.983) | 0.23 (5.446) | 5.12 (7.883) | -3.85 (5.868)
  Creatinine; Week2; n=41, 38, 14, 13 | -2.47 (7.966) | -2.78 (5.725) | 4.13 (6.518) | -1.17 (7.692)
  Creatinine; Week4; n=41, 39, 14, 13 | -3.4 (5.894) | -1.33 (6.403) | 5.35 (10.16) | -3.57 (9.599)
  Creatinine; Week6; n=41, 38, 13, 13 | -2.15 (6.18) | -0.34 (7.667) | 7.1 (7.905) | -2.05 (9.365)
  Creatinine; Week8; n=40, 39, 13, 13 | -1.88 (5.724) | -0.51 (5.425) | 9.43 (10.839) | -0.08 (10.23)
  Creatinine; Week12; n=38, 35, 12, 13 | -1.49 (8.411) | -1.99 (8.704) | 6.85 (10.363) | -2.41 (12.239)

13. Primary Outcome: Mean Change From Baseline in Chloride, Bicarbonate, Glucose, Potassium, Sodium, Inorganic Phosphorus and Urea/Blood Urea Nitrogen (BUN) at the Indicated Time Points up to Week 12
Description: Blood samples were collected for the measurement of Chloride, bicarbonate, glucose, potassium, sodium, inorganic phosphorus and urea/BUN at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4. Change from Baseline in the chloride, bicarbonate, glucose, potassium, sodium, inorganic phosphorus and urea/BUN values are summarized for each post-Baseline assessment until Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6, 8 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Millimoles per liter
  Chloride; Week1; n=40, 39, 15, 13 | 0.5 (2.1) | -0.4 (2.03) | 0.6 (2.61) | -0.2 (1.95)
  Chloride; Week2; n=41, 38, 14, 13 | 0.7 (2.37) | 0.1 (1.9) | 0.5 (1.61) | -0.7 (2.21)
  Chloride; Week4; n=41, 39, 14, 13 | 1.7 (2.31) | 1 (2.46) | 1.6 (2.21) | 0.1 (2.5)
  Chloride; Week6; n=41, 38, 13, 13 | 1.6 (2.62) | 0.8 (2.57) | 0.8 (2.73) | -0.1 (1.38)
  Chloride; Week8; n=40, 39, 13, 13 | 2 (3.49) | 0.7 (2.36) | 2.2 (3) | -0.8 (2.77)
  Chloride; Week12; n=37, 35, 12, 13 | 1.5 (2.36) | 0.1 (3.35) | 1.9 (2.61) | 1.2 (2.95)
  Bicarbonate; Week1; n=40, 39, 15, 13 | 0 (3.05) | -0.9 (2.57) | -1.2 (2.54) | -0.7 (2.56)
  Bicarbonate; Week2; n=41, 38, 14, 13 | -0.3 (2.2) | -0.8 (3.1) | -1.5 (2.98) | -0.2 (3.65)
  Bicarbonate; Week4; n=41, 39, 14, 13 | -0.9 (1.91) | -0.8 (2.55) | -1.4 (1.86) | -0.5 (2.67)
  Bicarbonate; Week6; n=41, 38, 13, 13 | -0.4 (2) | -0.7 (2.23) | -1.5 (2.18) | 0.6 (2.6)
  Bicarbonate; Week8; n=40, 39, 13, 13 | -0.7 (2.41) | -0.8 (2.35) | -1.2 (2.19) | 0 (2.2)
  Bicarbonate; Week12; n=37, 35, 12, 13 | -0.6 (2.42) | -0.9 (2.37) | -1.1 (2.23) | -0.5 (2.76)
  Glucose; Week1; n=40, 39, 15, 13 | -0.37 (1.485) | -0.34 (0.761) | -0.03 (0.616) | 0.36 (1.619)
  Glucose; Week2; n=41, 38, 14, 13 | -0.22 (1.467) | -0.17 (0.791) | 0.11 (0.52) | 0.13 (1.765)
  Glucose; Week4; n=41, 39, 14, 13 | -0.03 (1.162) | 0.02 (1.054) | -0.11 (0.601) | -0.48 (0.832)
  Glucose; Week6; n=41, 38, 13, 13 | -0.15 (1.315) | -0.18 (1.154) | 0.18 (0.772) | -0.55 (0.755)
  Glucose; Week8; n=40, 39, 13, 13 | -0.05 (1.165) | -0.06 (0.835) | 0.04 (0.675) | -0.36 (1.191)
  Glucose; Week12; n=38, 35, 12, 13 | -0.3 (1.877) | -0.39 (1.047) | -0.23 (0.757) | -0.45 (1.063)
  Potassium; Week1; n=40, 39, 15, 13 | -0.02 (0.392) | -0.06 (0.339) | -0.11 (0.376) | -0.02 (0.313)
  Potassium; Week2; n=41, 38, 14, 13 | -0.1 (0.428) | -0.12 (0.453) | -0.39 (0.417) | -0.02 (0.316)
  Potassium; Week4; n=41, 39, 14, 13 | -0.16 (0.411) | -0.11 (0.455) | -0.34 (0.497) | -0.05 (0.499)
  Potassium; Week6; n=41, 38, 13, 13 | -0.15 (0.483) | -0.16 (0.387) | -0.45 (0.355) | -0.21 (0.38)
  Potassium; Week8; n=40, 39, 13, 13 | -0.11 (0.49) | -0.19 (0.42) | -0.51 (0.348) | -0.14 (0.348)
  Potassium; Week12; n=37, 35, 12, 13 | -0.15 (0.394) | -0.21 (0.362) | -0.38 (0.447) | -0.1 (0.428)
  Sodium; Week1; n=40, 39, 15, 13 | -0.4 (1.85) | -0.8 (1.76) | -0.2 (2.46) | -0.8 (2.08)
  Sodium; Week2; n=41, 38, 14, 13 | -0.1 (2.15) | -0.6 (1.81) | 0 (1.8) | -1.3 (2.25)
  Sodium; Week4; n=41, 39, 14, 13 | 0.1 (2.16) | -0.1 (2.2) | 0.4 (1.78) | -0.8 (1.95)
  Sodium; Week6; n=41, 38, 13, 13 | 0.2 (2.39) | -0.3 (2.39) | 0.2 (2.91) | 0 (2)
  Sodium; Week8; n=40, 39, 13, 13 | 0.3 (3.28) | -0.6 (2.24) | 1.1 (2.18) | -0.6 (2.22)
  Sodium; Week12; n=37, 35, 12, 13 | 0.1 (1.91) | -0.3 (2.36) | 0.8 (2.66) | 0.5 (2.18)
  Inorganic Phosphorus; Week1; n=40, 39, 15, 13 | -0.13 (0.1599) | -0.086 (0.1415) | -0.122 (0.1353) | -0.087 (0.1489)
  Inorganic Phosphorus; Week2; n=41,38,14,13 | -0.141 (0.181) | -0.108 (0.1754) | -0.081 (0.1194) | -0.105 (0.1159)
  Inorganic Phosphorus; Week4; n=41,39,14,13 | -0.151 (0.1666) | -0.125 (0.1421) | -0.077 (0.1669) | -0.078 (0.1871)
  Inorganic Phosphorus; Week6; n=41,38,13,13 | -0.171 (0.1939) | -0.181 (0.1823) | -0.121 (0.1549) | -0.159 (0.121)
  Inorganic Phosphorus; Week8; n=40,39,13,13 | -0.169 (0.2025) | -0.23 (0.1937) | -0.112 (0.1563) | -0.14 (0.167)
  Inorganic Phosphorus; Week12; n=37,35,12,13 | -0.172 (0.1708) | -0.168 (0.2047) | -0.117 (0.1123) | -0.136 (0.1943)
  Urea/BUN; Week1; n=40, 39, 15, 13 | 0.24 (0.996) | 0.04 (1.002) | 0.19 (1.287) | -0.01 (1.188)
  Urea/BUN; Week2; n=41, 38, 14, 13 | 0.2 (1.012) | -0.13 (1.05) | 0.08 (1.309) | -0.12 (1.244)
  Urea/BUN; Week4; n=41, 39, 14, 13 | 0.03 (1.145) | -0.4 (1.047) | 0.11 (1.436) | -0.88 (1.137)
  Urea/BUN; Week6; n=41, 38, 13, 13 | -0.04 (1.09) | -0.29 (1.13) | -0.39 (0.883) | -1.02 (0.667)
  Urea/BUN; Week8; n=40, 39, 13, 13 | -0.16 (1.088) | -0.46 (1.337) | -0.07 (1.206) | -0.85 (1.067)
  Urea/BUN; Week12; n=37, 35, 12, 13 | -0.08 (1.164) | -0.31 (1.276) | -0.11 (1.272) | -0.64 (1.81)

14. Primary Outcome: Mean Change From Baseline in Creatinine Clearance at the Indicated Time Points up to Week 12
Description: Blood samples were collected for the measurement of Creatinine Clearance at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4. It is estimated by Cockcroft-Gault Equation. Change from Baseline in the Creatinine Clearance values are summarized for each post-Baseline assessment until Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6, 8 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milliliter per minute (mL/min)
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Milliliter per minute (mL/min)
  Creatinine Clearance; Week1; n=40, 39, 15, 13 | 1.5 (9.79) | -2.1 (19.51) | -9.5 (10.09) | 5.7 (10.18)
  Creatinine Clearance; Week2; n=41, 38,14,13 | 3.3 (13.48) | 4.7 (11.33) | -9 (12.55) | -1.8 (15.27)
  Creatinine Clearance; Week4; n=41, 39,14,13 | 5 (12.45) | 1.9 (14.72) | -9.1 (13.42) | 4.5 (16.19)
  Creatinine Clearance; Week6; n=41, 38,13,13 | 2.7 (11.93) | -0.7 (16.25) | -19.1 (20.54) | 1.5 (13.12)
  Creatinine Clearance; Week8; n=40, 39,13,13 | 1.9 (10.49) | 3.4 (19.94) | -17.8 (16.1) | -3 (14.54)
  Creatinine Clearance; Week12; n=38,35,12,13 | -0.2 (15.06) | 2.2 (17.27) | -14.3 (16.99) | 1.2 (20.49)

15. Primary Outcome: Number of Participants With Shift From Baseline in Urinalysis Data up to Week 12
Description: Urine samples were collected for urinalysis at Baseline, Weeks 2, 12, 18, 24, 48 and PT FU Weeks 4. Number of participants with shift from Baseline in urinalysis to normal (NL), abnormal (ANL) and missing (MIS) data up to Week 12 are summarized. Urine bilirubin (UBIL), urine glucose (UGLU), urine ketones (UKET), urine leukocyte esterase test (ULET) for detecting WBC, urine nitrite (UNIT), urine occult blood (UOB) were performed with dipstick method. Urine microscopy (UM) is performed to detect bacteria (BAC), red blood cells (RBC) and white blood cells (WBC). Other urinalysis parameter included urine pH (UpH) and urine specific gravity (USG). Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0), Weeks 2 and 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Participants
  Week 2, UBIL, BL MIS to PBL MIS, n=1,0,0,0 | 1 | 0 | 0 | 0
  Week 12, UBIL, BL MIS to PBL MIS,n=37,34,12,13 | 37 | 34 | 12 | 13
  Week 2, UGLU, BL MIS to PBL MIS, n=1,0,0,0 | 1 | 0 | 0 | 0
  Week 12, UGLU, BL MIS to PBL MIS,n=37,34,12,13 | 37 | 34 | 12 | 13
  Week 2, UKET, BL MIS to PBL MIS, n=1,0,0,0 | 1 | 0 | 0 | 0
  Week 12, UKET, BL MIS to PBL MIS,n=37,34,12,13 | 37 | 34 | 12 | 13
  Week 2, ULET, BL MIS to PBL MIS, n=1,0,0,0 | 1 | 0 | 0 | 0
  Week 12, ULET, BL MIS to PBL MIS,n=37,34,12,13 | 37 | 34 | 12 | 13
  Week 12, UMBT, BL MIS to PBL MIS,n=1,1,0,0 | 1 | 1 | 0 | 0
  Week 12, UMRBC, BL MIS to PBL MIS,n=4,5,2,2 | 4 | 5 | 2 | 2
  Week 12, UMWBC, BL MIS to PBL MIS, n=4,5,2,2 | 4 | 5 | 2 | 2
  Week 2, UNIT, BL MIS to PBL MIS, n=1,0,0,0 | 1 | 0 | 0 | 0
  Week 12, UNIT, BL MIS to PBL MIS,n=37,34,12,13 | 37 | 34 | 12 | 13
  Week 2, UOB, BL MIS to PBL MIS, n=1,0,0,0 | 1 | 0 | 0 | 0
  Week 12, UOB, BL MIS to PBL MIS,n=37,34,12,13 | 37 | 34 | 12 | 13
  Week 2, UPH, BL NL to PBL NL, n=1, 0,0,0 | 1 | 0 | 0 | 0
  Week 12, UPH, BL NL to PBL NL, n=37,34,12,13 | 36 | 34 | 12 | 13
  Week 12, UPH, BL NL to PBL ANL, n=37,34,12,13 | 1 | 0 | 0 | 0
  Week 2, USG, BL NL to PBL NL, n=1, 0,0,0 | 1 | 0 | 0 | 0
  Week 12, USG, BL NL to PBL NL, n=37,34,12,13 | 37 | 34 | 12 | 12
  Week 12, USG, BL NL to PBL ANL,n=37,34,12,13 | 0 | 0 | 0 | 1

16. Primary Outcome: Mean Change From Baseline in Electrocardiographic (ECG) Heart Rate Values at the Indicated Time Points up to Week 12
Description: The ECG parameter heart rate was measured at Baseline, Weeks 1 and 12. Change from Baseline in ECG heart rate is summarized for each post-Baseline assessment up to Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 1 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Beats per minute
  Week 1, n=41, 40, 15, 12 | 3.3 (8.28) | 0.8 (8.49) | 4.1 (9.52) | 4.8 (10.62)
  Week 12, n=38, 35, 12, 13 | 8.3 (8.37) | 5.1 (10.86) | 9.3 (10.15) | 8.5 (8)

17. Primary Outcome: Mean Change From Baseline in PR Interval, QRS Duration, Uncorrected QT Interval and QT Interval Corrected Bazett's Formula (QTcB), QT Interval Corrected Using Fridericia's Formula (QTcF) Values at the Indicated Time Points up to Week 12
Description: The ECG parameters including PR interval, QRS duration, uncorrected QT interval, QTcB, QTcF were measured at Baseline, Weeks 1 and 12. Change from Baseline in ECG parameters are summarized for each post-Baseline assessment up to Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 1 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Milliseconds
  PR interval, Week 1, n=41, 40, 15, 12 | 0.5 (19.43) | 1.2 (13.57) | 2.7 (7.27) | -1.6 (20.92)
  PR interval, Week 12, n=38, 35, 12, 13 | 2.9 (13.36) | 3.2 (12.07) | 5.5 (8.73) | 0.2 (14.68)
  QRS duration, Week 1, n=41, 40, 15,12 | -6.6 (50.28) | 0.4 (7.69) | 2.9 (6.61) | 0.4 (4.03)
  QRS duration, Week 12, n=38, 35, 12,13 | -8.2 (51.69) | -1.8 (6.44) | 0.4 (7.54) | -2 (4.4)
  Uncorrected QT Interval, Week 1, n=41,40,15,12 | -2.3 (27.29) | -2.6 (22.29) | -2.1 (22.39) | 5.9 (25.68)
  Uncorrected QT interval, Week 12,n=38,35,12,13 | -11.8 (31.28) | -12 (25.22) | -17 (18.01) | -4.6 (23.36)
  QTcB interval, Week 1, n=41,40,15,12 | 7.7087 (25.63001) | 0.2491 (22.90285) | 9.8112 (20.6771) | 19.8879 (40.13504)
  QTcB interval, Week 12,n=38,35,12,13 | 11.5512 (26.5644) | 1.7615 (20.3859) | 11.2801 (25.54652) | 18.9943 (16.76576)
  QTcF interval, Week 1, n=41,40,15,12 | 4.1995 (23.18239) | -0.7151 (19.69091) | 5.7676 (17.06472) | 14.9187 (32.2737)
  QTcF interval, Week 12,n=38,35,12,13 | 3.3516 (26.34546) | -3.1442 (17.38368) | 1.6147 (18.38188) | 10.7637 (17.07259)

18. Secondary Outcome: Number of Participants With Any AEs and Any SAEs After Week 12
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign(including an abnormal laboratory finding), symptom, or disease(new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, a congenital anomaly/birth defect, important medical events that jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition.
Time Frame: From Week 12 up to PT Week 24 FU
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Participants
  Any AE | 21 | 22 | 8 | 9
  Any SAE | 2 | 1 | 0 | 0

19. Secondary Outcome: Number of Participants Achieving Very Rapid Virologic Response (vRVR), Rapid Virologic Response (RVR), Complete Early Virologic Response (cEVR), Sustained Virologic Response 12 and 24 (SVR12 and SVR24) With Response Guided Treatment (RGT)
Description: Blood samples for the determination of HCV RNA levels were collected at Screening and Baseline, every study visit during the Treatment Period, and at PT FU Weeks 4, 12, and 24. vRVR is defined as plasma HCV RNA <LLOQ and target not detected 2 weeks after initiation of therapy. RVR is defined as plasma HCV RNA <LLOQ and target not detected 4 weeks after initiation of therapy. cEVR is defined as plasma HCV RNA <LLOQ and target not detected 12 weeks after initiation of therapy. SVR12 is defined as plasma HCV RNA <LLOQ and target not detected 12 weeks after completion of all therapy. SVR24 is defined as plasma HCV RNA <LLOQ and target not detected 24 weeks after completion of all therapy. SVR24 with RGT are participants who achieved both SVR24 and eRVR.
Time Frame: From the start of the treatment up to PT FU Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Participants
  vRVR | 8 | 12 | 8 | 6
  RVR | 23 | 23 | 10 | 9
  cEVR | 33 | 30 | 11 | 13
  SVR12 | 30 | 26 | 10 | 0
  SVR24 | 27 | 25 | 10 | 0
  SVR24 with RGT | 17 | 17 | 9 | 0

20. Secondary Outcome: Mean GSK2336805 Plasma Concentrations on Day 1, Day 2, Week 4, and Week 12
Description: Plasma pharmacokinetic (PK) samples were collected for all participants on Day 1 (0 hour [h]-1h, 1h-4h, 4h-8h, 8h-20h), Day 2 (Predose [20-28h]), Week 4 (Predose [20-28h], 0h-1h, 1h-4h, 4h-8h, 8h-20h, 20h-28h) and Week 12 (Predose [20-28h]). PK Population is comprised of all participants who received GSK2336805 and underwent plasma PK sampling (intensive or sparse) during the study.
Time Frame: Day 1, Day 2, Week 4, and Week 12
Population: PK Population included all participants who received GSK2336805 and underwent plasma PK sampling (intensive or sparse) during the study. Only participants for whom plasma PK samples were obtained were assessed (represented by n=X, X in category titles).
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV: Participants with chronic G1 and G4 HCV infection received GSK2336805 60 mg orally (30 mg x 2tablets) once daily in the morning with food in combination with antiviral therapy (PEG+RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was180 µg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if bodyweight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken orally in 2divided doses with food.
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV
Number analyzed (Participants) | 41 | 53
nanograms per milliliter (ng/mL)
  Day 1 (0h-1h), n=1, 3 | NA (NA) — A value of NA indicates not applicable | 604 (392.763)
  Day 1 (1h-4h), n=35, 42 | 290.39 (241.05) | 445.18 (314.624)
  Day 1 (4h-8h), n=0, 3 | NA (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | 221.33 (191.996)
  Day 1 (8h-20h), n=0, 1 | NA (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | NA (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation).
  Day 2 Predose (20-28h), n=36, 43 | 53.79 (52.629) | 123.89 (257.575)
  Week 4 Predose (20-28h), n=33, 42 | 81.18 (153.462) | 146.85 (243.331)
  Week 4 (0h-1h), n=2, 6 | 198.4 (242.679) | 553 (536.451)
  Week 4 (1h-4h), n=46, 52 | 392.78 (275.504) | 591.07 (402.442)
  Week 4 (4h-8h), n=22, 19 | 215.55 (127.737) | 411.68 (251.604)
  Week 4 (8h-20h), n=1, 2 | NA (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | 192.5 (94.045)
  Week 4 (20h-28h), n=11, 10 | 51.24 (57.261) | 66.29 (53.604)
  Week 12 (Predose [20-28h]), n=26, 35 | 45.99 (42.034) | 142.59 (178.252)

21. Secondary Outcome: Maximum Plasma Concentration (Cmax) and Concentration at the End of the Dosing Interval (Ctau) of GSK2336805 at Week 4
Description: Blood samples for PK analysis of GSK2336805 was obtained on Week 4+1 day at predose and at 1, 2, 4, 7, 24 hours post-dose.
Time Frame: Week 4 (24 h post dose)
Population: Intensive PK Summary Population: Intensive PK Summary Population comprised of participants with evaluable GSK2336805 PK parameters at Week 4. Only participants available at the indicated time point were assessed (represented by n=X, X in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV: Participants with chronic G1 and G4 HCV infection received GSK2336805 60 mg orally (30 mg x 2tablets) OD in the morning with food in combination with antiviral therapy (PEG+RIBA) for 12 weeksfollowed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was180 μg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if bodyweight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken orally in 2divided doses with food.
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV
Number analyzed (Participants) | 11 | 10
ng/mL
  Cmax, n=11, 10 | 335.35 (69.4) | 618.75 (46.1)
  Ctau, n=11, 10 | 31.37 (135.9) | 49.31 (97.6)

22. Secondary Outcome: Time of Maximal Plasma Concentration (Tmax) of GSK2336805 at Week 4
Description: Blood samples for PK analysis of GSK2336805 was obtained on Week 4+1 day at predose and at 1, 2, 4, 7, 24 hours postdose.
Time Frame: Week 4 (24 h post dose)
Population: Intensive PK Summary Population
Measure: Median (Full Range); unit: hour
Groups:
- GSK2336805 40 mg, Genotype 1 HCV: Participants with chronic G1 HCV infection received GSK2336805 40 mg orally (20 mg x 2 tablets) once daily in the morning with food in combination with antiviral therapy (PEG + RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on the eRVR achievement. PEG dose was 180 ug once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight is <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight is >=75 kg) taken in 2 divided doses with food.
- GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV: Participants with chronic G1 and G4 HCV infection received GSK2336805 60 mg orally (30 mg x 2tablets) OD in the morning with food in combination with antiviral therapy (PEG+RIBA) for 12 weeksfollowed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was180 μg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if bodyweight is <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight is >=75 kg) taken orally in 2divided doses with food.
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV
Number analyzed (Participants) | 11 | 10
hour | 2 [1 to 4] | 2 [1 to 7]

23. Secondary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUC[0-tau]) at Week 4
Description: Blood samples for PK analysis of GSK2336805 was obtained on Week 4+1 day at predose and at 1, 2, 4, 7 and 24 hours postdose.
Time Frame: Week 4 (24 h post dose)
Population: Intensive PK Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter(hr*ng/mL)
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV
Number analyzed (Participants) | 11 | 10
hour*nanogram per milliliter(hr*ng/mL) | 2733.34 (82) | 4948.23 (66.3)

24. Secondary Outcome: Apparent Clearance (CL/F) at Week 4
Description: Blood samples for PK analysis of GSK2336805 was obtained on Week 4+1 day at predose and at 1, 2, 4, 7 and 24 hours postdose. CL/F was calculated as dose divided by AUC(0-tau).
Time Frame: Week 4 (24 h post dose)
Population: Intensive PK Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV
Number analyzed (Participants) | 11 | 10
Liter per hour (L/hr) | 14.63 (82) | 12.13 (66.3)

25. Secondary Outcome: Apparent Volume of Distribution (Vz/F) at Week 4
Description: Blood samples for PK analysis of GSK2336805 was obtained on Week 4+1 day at predose and at 1, 2, 4, 7 and 24 hours postdose. Vz/F was calculated as dose divided by (AUC[0-tau] lambda z) where lambda z is the terminal phase rate constant.
Time Frame: Week 4 (24 h post dose)
Population: Intensive PK Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV
Number analyzed (Participants) | 11 | 10
Liter per hour (L/hr) | 172.81 (76.6) | 125.09 (67.9)

26. Secondary Outcome: Mean Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count and White Blood Cell Count at the Indicated Time Points After Week 12
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelet count and white blood cell count at the Baseline, Day 2, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT Week 4. Change from Baseline in the basophils, eosinophils, lymphocytes, total neutrophils platelet count and white blood cell count values are summarized for each post-Baseline assessment after Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Giga cells per liter
  Basophils; Week18; n=37, 33, 13, 12 | -0.019 (0.0178) | -0.01 (0.0194) | -0.014 (0.0112) | -0.012 (0.0119)
  Basophils; Week24; n=34, 32, 12, 11 | -0.018 (0.0177) | -0.01 (0.0166) | -0.013 (0.0129) | -0.013 (0.011)
  Basophils; Week30; n=13, 10, 2, 2 | -0.018 (0.0142) | -0.012 (0.0148) | -0.02 (0) | -0.02 (0)
  Basophils; Week36; n=12, 7, 1, 2 | -0.02 (0.0165) | -0.006 (0.019) | -0.02 (NA) — A value of NA indicates not applicable | -0.01 (0.0141)
  Basophils; Week42; n=10, 6, 2, 2 | -0.015 (0.0242) | -0.005 (0.0187) | 0 (0.0424) | -0.015 (0.0071)
  Basophils; Week48; n=7, 6, 1, 2 | -0.007 (0.0214) | -0.007 (0.0197) | 0.02 (NA) — System value of NA indicates not applicable (too few participants). | 0.005 (0.0071)
  Basophils; PT Week4; n=32, 34, 11, 11 | -0.007 (0.0162) | -0.003 (0.0189) | -0.001 (0.0181) | -0.003 (0.0119)
  Eosinophils; Week18; n=37, 33, 13, 12 | -0.119 (0.1006) | -0.127 (0.1207) | -0.087 (0.0507) | -0.068 (0.0746)
  Eosinophils; Week24; n=34, 32, 12, 11 | -0.128 (0.101) | -0.131 (0.1103) | -0.118 (0.0612) | -0.041 (0.1003)
  Eosinophils; Week30; n=13, 10, 2, 2 | -0.124 (0.0982) | -0.116 (0.1117) | -0.13 (0.0849) | -0.04 (0.0141)
  Eosinophils; Week36; n=12, 7, 1, 2 | -0.081 (0.1459) | -0.123 (0.1003) | -0.06 (NA) — System value of NA indicates not applicable (too few participants). | -0.05 (0.0141)
  Eosinophils; Week42; n=10, 6, 2, 2 | -0.105 (0.074) | -0.1 (0.12) | -0.02 (0.0424) | -0.04 (0)
  Eosinophils; Week48; n=8, 6, 1, 2 | -0.071 (0.0889) | -0.11 (0.1223) | 0.13 (NA) — System value of NA indicates not applicable (too few participants). | -0.05 (0.0141)
  Eosinophils; PT Week4; n=32, 34, 11,11 | -0.069 (0.0925) | -0.085 (0.1208) | -0.07 (0.0694) | -0.018 (0.0808)
  Lymphocytes; Week18; n=37, 33, 13,12 | -1.081 (0.5533) | -1.157 (0.5373) | -0.999 (0.4672) | -0.973 (0.5328)
  Lymphocytes; Week24; n=34, 32, 12,11 | -1.181 (0.4795) | -1.092 (0.5598) | -1.405 (0.5912) | -1.057 (0.4832)
  Lymphocytes; Week30; n=13, 10, 2, 2 | -1.225 (0.7588) | -1.085 (0.798) | -1.905 (0.1768) | -1.845 (0.2899)
  Lymphocytes; Week36; n=12, 7, 1, 2 | -1.267 (0.6828) | -1.286 (0.8983) | -1.97 (NA) — System value of NA indicates not applicable (too few participants). | -1.92 (0.4808)
  Lymphocytes; Week42; n=10, 6, 2, 2 | -1.135 (0.8657) | -1.22 (0.9909) | -1.125 (1.0253) | -1.93 (0.1414)
  Lymphocytes; Week48; n=7, 6, 1, 2 | -0.779 (1.0639) | -1.4 (1.0384) | 0.09 (NA) — System value of NA indicates not applicable (too few participants). | -2.2 (0.0424)
  Lymphocytes; PT Week4; n=32, 34, 11,11 | -0.681 (0.4594) | -0.7 (0.6163) | -0.756 (0.5874) | -0.737 (0.5666)
  Monocytes; Week18; n=37, 33, 13, 12 | -0.186 (0.1588) | -0.141 (0.1339) | -0.088 (0.1663) | -0.143 (0.1776)
  Monocytes; Week24; n=34, 32, 12, 11 | -0.206 (0.1692) | -0.156 (0.1574) | -0.151 (0.1474) | -0.121 (0.1902)
  Monocytes; Week30; n=13, 10, 2, 2 | -0.151 (0.1655) | -0.135 (0.091) | -0.4 (0.3111) | -0.06 (0.0141)
  Monocytes; Week36; n=12, 7, 1, 2 | -0.255 (0.1474) | -0.18 (0.0987) | -0.2 (NA) — System value of NA indicates not applicable (too few participants). | 0.015 (0.1061)
  Monocytes; Week42; n=10, 6, 2, 2 | -0.184 (0.234) | -0.093 (0.1743) | -0.025 (0.2192) | -0.01 (0.099)
  Monocytes; Week48; n=7, 6, 1, 2 | -0.066 (0.1744) | -0.147 (0.088) | 0.02 (NA) — System value of NA indicates not applicable (too few participants). | -0.085 (0.1909)
  Monocytes; PT Week4; n=32, 34, 11,11 | -0.047 (0.1773) | -0.031 (0.165) | 0.032 (0.1543) | -0.053 (0.1536)
  Total Neutrophils; Week18; n=37, 33,13,12 | -2.702 (1.9136) | -2.378 (1.6735) | -1.652 (0.852) | -1.463 (0.7174)
  Total Neutrophils; Week24; n=34, 32,12,11 | -2.527 (1.9492) | -2.187 (1.7758) | -1.308 (0.7148) | -1.3 (0.9956)
  Total Neutrophils; Week30; n=13, 10,2,2 | -2.402 (1.7954) | -2.252 (2.3658) | -2.24 (1.2869) | -2.085 (0.1909)
  Total Neutrophils; Week36; n=12, 7, 1,2 | -2.503 (1.6709) | -2.777 (2.4215) | -1.61 (NA) — System value of NA indicates not applicable (too few participants). | -1.63 (0.297)
  Total Neutrophils; Week42; n=10, 6, 2,2 | -2.23 (2.0311) | -3.085 (2.7313) | -0.565 (0.7849) | -1.815 (0.4455)
  Total Neutrophils; Week48; n=7, 6, 1, 2 | -1.129 (2.2597) | -2.488 (3.397) | 0.02 (NA) — System value of NA indicates not applicable (too few participants). | -1.445 (0.4596)
  Total Neutrophils; PT Week4; n=32, 34,11,11 | -1.158 (1.8855) | -0.808 (1.6104) | -0.744 (1.1276) | -0.671 (0.8001)
  Platelet Count; Week18; n=38, 34, 13,12 | -73.7 (43.93) | -87.5 (38.4) | -55.7 (56.96) | -52.1 (39.87)
  Platelet Count; Week24; n=35, 33, 12,11 | -67.5 (43.22) | -78.8 (44.15) | -60.3 (56.5) | -51.9 (44.19)
  Platelet Count; Week30; n=13, 10, 1, 2 | -70 (60.5) | -71.9 (59.35) | -112 (NA) — System value of NA indicates not applicable (too few participants). | -36.5 (47.38)
  Platelet Count; Week36; n=12, 7, 1, 2 | -64.1 (41.52) | -75.7 (65.89) | -115 (NA) — System value of NA indicates not applicable (too few participants). | -34 (52.33)
  Platelet Count; Week42; n=10, 6, 2, 2 | -56.1 (53.01) | -67.3 (62.09) | -112 (0) | -22 (52.33)
  Platelet Count; Week48; n=9, 6, 1, 2 | -37.7 (66.18) | -68.8 (65.74) | 33 (NA) — System value of NA indicates not applicable (too few participants). | -14 (22.63)
  Platelet Count; PT Week4; n=32, 34,11,11 | -20.4 (44.37) | -28.9 (45.92) | -12.4 (34.3) | -12.9 (42.3)
  White Blood Cell count; Week18; n=37,33,13,12 | -4.1 (2.258) | -3.81 (1.884) | -2.84 (0.961) | -2.65 (0.923)
  White Blood Cell count ; Week24; n=34,32,12,11 | -4.06 (2.251) | -3.58 (1.977) | -3 (1.047) | -2.52 (1.272)
  White Blood Cell count ; Week30; n=13,10,2,2 | -3.92 (2.258) | -3.59 (3.051) | -4.7 (1.838) | -4.05 (0.495)
  White Blood Cell count ; Week36; n=12,7,1,2 | -4.13 (2.188) | -4.39 (3.168) | -3.9 (NA) — System value of NA indicates not applicable (too few participants). | -3.55 (0.919)
  White Blood Cell count ; Week42; n=10,6,2,2 | -3.67 (2.807) | -4.52 (3.68) | -1.75 (2.051) | -3.8 (0.707)
  White Blood Cell count; Week48; n=7,6,1,2 | -2.09 (3.304) | -4.17 (4.172) | 0.2 (NA) — System value of NA indicates not applicable (too few participants). | -3.8 (0.141)
  White Blood Cell count; PT Week4;n=32,34,11,11 | -1.97 (1.938) | -1.64 (1.907) | -1.54 (1.638) | -1.45 (0.884)

27. Secondary Outcome: Mean Change From Baseline in Red Blood Cell Count at the Indicated Time Points After Week 12
Description: Blood samples were collected for the measurement of red blood cell count at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Week 4. Change from Baseline in the red blood cell count values are summarized for each post-Baseline assessment after Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Trillion cells per liter
  Red Blood Cell count; Week 18; n=38, 34, 13, 12 | -1.13 (0.494) | -0.88 (0.591) | -1.19 (0.638) | -0.99 (0.498)
  Red Blood Cell count; Week 24; n=35, 33, 12, 11 | -1.13 (0.482) | -0.94 (0.513) | -1.19 (0.552) | -1.14 (0.528)
  Red Blood Cell count; Week 30; n=13,10,2,2 | -1.05 (0.511) | -0.75 (0.809) | -1.45 (0.071) | -1.45 (0.354)
  Red Blood Cell count; Week 36; n=12,7,1,2 | -0.88 (0.67) | -1.06 (0.761) | -1 (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | -1.3 (0.283)
  Red Blood Cell count; Week 42; n=10,6,2,2 | -0.91 (0.674) | -1.17 (0.769) | -0.55 (0.636) | -1.45 (0.354)
  Red Blood Cell count; Week 48; n=9, 6,1,2 | -0.83 (0.791) | -1.03 (0.794) | -0.4 (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | -1.5 (0.566)
  Red Blood Cell count; PT Week 4; n=32,34,11,11 | -0.57 (0.435) | -0.37 (0.353) | -0.66 (0.437) | -0.65 (0.474)

28. Secondary Outcome: Mean Change From Baseline in Hemoglobin at the Indicated Time Points After Week 12
Description: Blood samples were collected for the measurement of hemoglobin at the the Baseline, Day 2, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Week 4. Change from Baseline in the hemoglobin values are summarized for each post-Baseline assessment after Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Grams per liter
  Hemoglobin; Week 18; n=38, 34, 13, 12 | -33.6 (12.34) | -26.7 (14.65) | -35 (16.38) | -29 (10.61)
  Hemoglobin; Week 24; n=35, 33, 12,11 | -33.4 (12.16) | -28 (12.44) | -35.6 (13.48) | -32.3 (14.98)
  Hemoglobin; Week 30; n=13, 10, 2, 2 | -30.2 (16.13) | -21 (20.02) | -40 (12.73) | -40 (1.41)
  Hemoglobin; Week 36; n=12, 7, 1, 2 | -26.7 (18.86) | -30 (16.37) | -37 (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | -35 (1.41)
  Hemoglobin; Week 42; n=10, 6, 2, 2 | -27.1 (18.51) | -31.7 (19.82) | -25 (22.63) | -40 (1.41)
  Hemoglobin; Week 48; n=9, 6, 1, 2 | -25.9 (21.47) | -29.3 (20.33) | -18 (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | -41 (8.49)
  Hemoglobin; PT Week 4; n=32, 34, 11,11 | -16.5 (11.43) | -11.7 (9.57) | -21.4 (8.59) | -16.8 (11.99)

29. Secondary Outcome: Mean Change From Baseline in Hematocrit at the Indicated Time Points After Week 12
Description: Blood samples were collected for the measurement of hematocrit at the the Baseline, Day 2, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Week 4. Change from Baseline in the hematocrit values are summarized for each post-Baseline assessment after Week 12. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Ratio
  Hematocrit; Week 18; n=38, 34, 13, 12 | -0.083 (0.03831) | -0.0622 (0.04289) | -0.0776 (0.04313) | -0.0699 (0.02801)
  Hematocrit; Week 24; n=35, 33, 12, 11 | -0.0782 (0.04021) | -0.0635 (0.03499) | -0.0808 (0.03543) | -0.0823 (0.03968)
  Hematocrit; Week 30; n=13, 10, 2, 2 | -0.0713 (0.0486) | -0.0397 (0.05793) | -0.0955 (0.03323) | -0.1125 (0.00636)
  Hematocrit; Week 36; n=12, 7, 1, 2 | -0.0567 (0.05031) | -0.069 (0.04724) | -0.087 (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable). | -0.0895 (0.00354)
  Hematocrit; Week 42; n=10, 6, 2, 2 | -0.0623 (0.05449) | -0.0802 (0.0562) | -0.0535 (0.07) | -0.111 (0.00566)
  Hematocrit; Week 48; n=9, 6, 1, 2 | -0.0624 (0.06203) | -0.0753 (0.05285) | -0.047 (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable). | -0.1095 (0.03041)
  Hematocrit; PT Week 4; n=32, 34, 11,11 | -0.0293 (0.03575) | -0.0135 (0.03178) | -0.0362 (0.02907) | -0.0354 (0.0358)

30. Secondary Outcome: Mean Change From Baseline in Mean Corpuscle Volume at the Indicated Time Points After Week 12
Description: Blood samples were collected for the measurement of mean corpuscle volume at the the Baseline, Day 2, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Week 4. Change from Baseline in the mean corpuscle volume values are summarized for each post-Baseline assessment after Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Femtoliters
  Mean Corpuscle Volume ; Week 18;n=38,34,13,12 | 7.5 (6.37) | 6.2 (8.19) | 8.5 (5.78) | 5.3 (5.28)
  Mean Corpuscle Volume ; Week 24;n=35,33,12,11 | 8.5 (6.14) | 7.5 (8.89) | 7.6 (5.9) | 5.8 (5.08)
  Mean Corpuscle Volume ; Week 30; n=13,10,2,2 | 7.8 (7.24) | 9.5 (12.02) | 11.5 (7.78) | 3 (2.83)
  Mean Corpuscle Volume ; Week 36; n=12,7,1,2 | 8.1 (5.92) | 11.4 (13.6) | 2 (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | 5.5 (2.12)
  Mean Corpuscle Volume ; Week 42;n=10,6,2,2 | 6.9 (5.7) | 10.7 (14.47) | 1 (2.83) | 4 (2.83)
  Mean Corpuscle Volume ; Week 48;n=9,6,1,2 | 5.2 (5.76) | 9 (14.04) | -1 (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | 5 (1.41)
  Mean Corpuscle Volume; PT Week 4; n=32,34,11,11 | 6.1 (5.56) | 5.1 (4.86) | 5.8 (3.79) | 5.3 (5.1)

31. Secondary Outcome: Mean Change From Baseline in Albumin at the Indicated Time Points After Week 12
Description: Blood samples were collected for the measurement of albumin at the the Baseline, Day 2, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Week 4. Change from Baseline in the albumin values are summarized for each post-Baseline assessment after Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Grams per liter
  Albumin; Week 18; n=38, 34, 13, 12 | -2.3 (2.78) | -1.4 (2.65) | -1.8 (2.86) | -1 (2.89)
  Albumin; Week 24; n=35, 33, 12, 11 | -2.1 (3.08) | -1.6 (2.82) | -2.3 (2.81) | -1.1 (2.81)
  Albumin; Week 30; n=13, 10, 3, 2 | -1.8 (2.09) | -0.7 (4.22) | -3 (2.65) | -4.5 (0.71)
  Albumin; Week 36; n=10, 7, 2, 2 | -1.7 (3.92) | -1.1 (2.85) | 2 (1.41) | -2 (0)
  Albumin; Week 42; n=9, 6, 1, 2 | -1.3 (2.5) | -1.3 (1.63) | -1 (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | -3 (0)
  Albumin; Week 48; n=6, 6, 0, 2 | -1.3 (3.61) | -0.3 (2.16) | NA (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | -4 (1.41)
  Albumin; PT Week 4; n=33, 34, 11, 11 | -0.7 (3.93) | -0.2 (2.84) | 0.5 (2.3) | -0.7 (1.79)

32. Secondary Outcome: Mean Change From Baseline in ALP, ALT, AST, CK and GGT at the Indicated Time Points After Week 12
Description: Blood samples were collected for the measurement of ALP, ALT, AST, CK and GGT at the the Baseline, Day 2, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Week 4. Change from Baseline in the ALP, ALT, AST, CK and GGT values are summarized for each post-Baseline assessment after Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International units per liter
Groups:
- GSK2336805 60 mg, Genotype 1 HCV: Participants with chronic G1 HCV infection received GSK2336805 60 mg orally (30 mg x 2 tablets) once daily in the morning with food in combination with antiviral therapy (PEG+RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was 180 µg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight is >=75 kg) taken orally in 2 divided doses with food.
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
International units per liter
  ALP; Week 18; n=38, 34, 13, 12 | 2.5 (17.25) | 1.1 (16.95) | 2.2 (21.77) | 6.4 (20.08)
  ALP; Week 24; n=35, 33, 12, 11 | 0.8 (19.71) | 3.3 (18.83) | 2.1 (20.24) | 4.5 (22.82)
  ALP; Week 30; n=13, 10, 3, 2 | 1.8 (15.79) | -6.4 (18.62) | -8 (8.54) | 22.5 (14.85)
  ALP; Week 36; n=10, 7, 2, 2 | 2 (17.49) | 2.7 (9.45) | 2.5 (0.71) | 18 (7.07)
  ALP; Week 42; n=9, 6, 1, 2 | 5.3 (13.4) | 3.3 (8.45) | -2 (NA) — System value of NA indicates not applicable (too few participants). | 17.5 (2.12)
  ALP; Week 48; n=6, 6, 0, 2 | 9.8 (17.36) | 4.2 (9.62) | NA (NA) — System value of NA indicates not applicable (too few participants). | 30 (24.04)
  ALP; PT Week 4; n=33, 34, 11, 11 | -4.9 (19.71) | -6.3 (17.88) | -7 (17.93) | -3.9 (22.15)
  ALT; Week 18; n=38, 34, 13, 12 | -38.9 (61.39) | -22.9 (61.65) | -38.6 (40.89) | -38.4 (32.63)
  ALT; Week 24; n=35, 33, 12, 11 | -43.9 (62.25) | -31.3 (56.12) | -39.7 (38.19) | -41.7 (28.32)
  ALT; Week 30; n=13, 10, 3, 2 | -34.8 (30.82) | -45.1 (95.76) | -57.7 (58.31) | -26 (22.63)
  ALT; Week 36; n=10, 7, 2, 2 | -30.2 (28.15) | -16.6 (13.7) | -69 (74.95) | -20.5 (16.26)
  ALT; Week 42; n=9, 6, 1, 2 | -34.3 (35.15) | -14.3 (20.07) | -122 (NA) — System value of NA indicates not applicable (too few participants). | -28 (25.46)
  ALT; Week 48; n=6, 6, 0, 2 | -38.8 (42.1) | -10.8 (27.11) | NA (NA) — System value of NA indicates not applicable (too few participants). | -26.5 (26.16)
  ALT; PT Week 4; n=33, 34, 11, 11 | -45.5 (62.76) | -33.3 (56.81) | -31.5 (22.68) | -43.9 (27.71)
  AST; Week 18; n=38, 34, 13, 12 | -13.1 (27.49) | -3.5 (37.25) | -18.8 (27.32) | -16.3 (15.11)
  AST; Week 24; n=35, 33, 12, 11 | -16.5 (26.86) | -11.8 (30.51) | -23.8 (26.91) | -15.7 (18.91)
  AST; Week 30; n=13, 10, 3, 2 | -15.1 (17.35) | -18.7 (43.89) | -27.7 (20.13) | -6.5 (7.78)
  AST; Week 36; n=10, 7, 2, 2 | -11.8 (13.81) | -7.3 (9.5) | -27.5 (31.82) | -2.5 (2.12)
  AST; Week 42; n=9, 6, 1, 2 | -14.2 (16.81) | -5.8 (10.03) | -54 (NA) — System value of NA indicates not applicable (too few participants). | -9 (7.07)
  AST; Week 48; n=6, 6, 0, 2 | -12.8 (18.65) | -2.2 (13.61) | NA (NA) — System value of NA indicates not applicable (too few participants). | -6.5 (9.19)
  AST; PT Week 4; n=33, 34, 11, 11 | -19.5 (26.41) | -15.6 (34.38) | -17.7 (14.67) | -16 (31.8)
  CK; Week 18; n=38, 34, 13, 12 | -44 (55.77) | -28.3 (36.59) | -38.7 (45.46) | -60.7 (75.8)
  CK; Week 24; n=35, 33, 12, 11 | -34.5 (66.48) | -18.7 (77.24) | -39 (36.68) | 60.1 (475.39)
  CK; Week 30; n=13, 10, 3, 2 | -33 (83.25) | -15.8 (51.92) | -30 (24.27) | -78.5 (55.86)
  CK; Week 36; n=10, 7, 2, 2 | -18.9 (34.18) | -26.7 (32.22) | -37.5 (6.36) | -69 (53.74)
  CK; Week 42; n=9, 6, 1, 2 | -0.2 (51.5) | -29.7 (43.42) | -32 (NA) — System value of NA indicates not applicable (too few participants). | -81 (57.98)
  CK; Week 48; n=6, 6, 0, 2 | 10.5 (71.39) | 22.3 (77.32) | NA (NA) — System value of NA indicates not applicable (too few participants). | -82.5 (70)
  CK; PT Week 4; n=33, 34, 11, 11 | -17.9 (48.82) | -26.4 (49.42) | -21.7 (42.62) | 258.7 (994.88)
  GGT; Week 18; n=38, 34, 13, 12 | -37.3 (71.19) | -12.3 (60.35) | -30.2 (42.04) | -34.2 (56.52)
  GGT; Week 24; n=35, 33, 12, 11 | -38.3 (72.79) | -12.5 (86.73) | -37.4 (45.44) | -35.7 (59.63)
  GGT; Week 30; n=13, 10, 3, 2 | -44.2 (41.3) | -32.8 (31.81) | -38.7 (36.02) | -12 (4.24)
  GGT; Week 36; n=10, 7, 2, 2 | -51.5 (45.03) | -19.7 (24.52) | -40.5 (33.23) | -10 (4.24)
  GGT; Week 42; n=9, 6, 1, 2 | -44.6 (46.61) | -19.7 (25.06) | -17 (NA) — System value of NA indicates not applicable (too few participants). | -9 (1.41)
  GGT; Week 48; n=6, 6, 0, 2 | -37.8 (28.74) | -16.8 (24.38) | NA (NA) — System value of NA indicates not applicable (too few participants). | -9.5 (6.36)
  GGT; PT Week 4; n=33, 34, 11, 11 | -43.4 (78.29) | -17.7 (78.22) | -30.7 (41.91) | -41.4 (61.06)

33. Secondary Outcome: Mean Change From Baseline in Total Bilirubin and Creatinine at the Indicated Time Points After Week 12
Description: Blood samples were collected for the measurement of total bilirubin and creatinine at the the Baseline, Day 2, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Week 4. Change from Baseline in the direct bilirubin, total bilirubin and creatinine values are summarized for each post-Baseline assessment afterl Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Micromoles per liter
  Total bilirubin; Week 18; n=38, 34, 13, 12 | 0.5 (5.01) | 1.7 (5.32) | -1.4 (11.37) | 0.6 (6.49)
  Total bilirubin; Week 24; n=35, 33, 12,11 | -0.1 (5.73) | 1 (4.08) | -1.3 (11.9) | 1.3 (6.26)
  Total bilirubin; Week 30; n=13, 10, 3, 2 | -0.2 (5.99) | 0.8 (4.76) | -2.3 (9.29) | -4 (5.66)
  Total bilirubin; Week 36; n=10, 7, 2, 2 | 0 (4.29) | 1.9 (4.95) | -3 (11.31) | -3 (7.07)
  Total bilirubin; Week 42; n=9, 6, 1, 2 | 0.1 (5.11) | 1.5 (5.79) | -14 (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | -4 (5.66)
  Total bilirubin; Week 48; n=6, 6, 0, 2 | -0.7 (4.72) | 3.5 (7.2) | NA (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | -4 (2.83)
  Total bilirubin PT Week 4; n=33, 34, 11,11 | -4.6 (3.57) | -2.4 (3.3) | -0.4 (5.68) | -2.2 (2.71)
  Creatinine; Week 24; n=35, 33, 12, 11 | -1.55 (9.507) | -2.4 (8.413) | -3.12 (9.408) | 1.31 (10.377)
  Creatinine; Week 18; n=38, 34, 13, 12 | -2.24 (9.186) | -1.97 (9.65) | -1.75 (9.874) | 0.09 (10.668)
  Creatinine; Week 30; n=13, 10, 3, 2 | 0.66 (4.603) | 2.82 (8.123) | -8.47 (8.693) | -8.85 (3.748)
  Creatinine; Week 36; n=10, 7, 2, 2 | 2.33 (11.096) | 2.99 (8.179) | -5.5 (16.829) | -8 (1.273)
  Creatinine; Week 42; n=9, 6, 1, 2 | 1.23 (10.32) | 4.97 (11.697) | -14.3 (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | -7.55 (5.586)
  Creatinine; Week 48; n=6, 6, 0, 2 | -2.35 (4.222) | 10.07 (17.173) | NA (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | -7.1 (1.273)
  Creatinine; PT Week 4; n=33, 34, 11,11 | 1.23 (8.22) | -0.34 (7.624) | -1.7 (6.897) | -1.25 (6.228)

34. Secondary Outcome: Mean Change From Baseline in SBP and DBP at the Indicated Time Points After Week 12
Description: Blood pressure measurements were taken to observe vital signs and included SBP and DBP at the Baseline, Day 2, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4. As defined in the Reporting Analysis Plan (RAP) for this protocol, the supplemental final data package generated for this study after Week 12 only provided graphical displays of vital signs (e.g., change from baseline for heart rate and blood pressure) to facilitate clinical interpretation and data summarization. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed. All abnormal values and statistical summary tables were not available after week 12.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: Safety Population
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 0 | 0 | 0 | 0

35. Secondary Outcome: Mean Change From Baseline in Heart Rate at the Indicated Time Points After Week 12
Description: Vital sign monitoring included heart rate, measured at the Baseline, Day 2, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4. As defined in the Reporting Analysis Plan (RAP) for this protocol, the supplemental final data package generated for this study after Week 12 only provided graphical displays of vital signs (e.g., change from Baseline for heart rate and blood pressure) to facilitate clinical interpretation and data summarization. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed. All abnormal values and statistical summary tables were not available after week 12.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: Safety Population
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 0 | 0 | 0 | 0

36. Secondary Outcome: Mean Change From Baseline in ECG Heart Rate Values at the Indicated Time Points After Week 12
Description: The ECG data was only collected "Perform as needed", therefore, no such summary table was generated. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: Safety Population
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 0 | 0 | 0 | 0

37. Secondary Outcome: Mean Change From Baseline in PR Interval, QRS Duration, Uncorrected QT Interval, QTcB, QTcF Values at the Indicated Time Points After Week 12
Description: as for outcome 36
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: Safety Population
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 0 | 0 | 0 | 0

38. Secondary Outcome: Mean Change From Baseline in Chloride, Bicarbonate, Glucose, Potassium, Sodium, Inorganic Phosphorus and Urea/BUN at the Indicated Time Points After Week 12
Description: Blood samples were collected for the measurement of Chloride, bicarbonate, glucose, potassium, sodium, inorganic phosphorus and urea/bun at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4. Change from Baseline in the Chloride, Bicarbonate, Glucose, Potassium, Sodium, Inorganic Phosphorus and Urea/Bun values are summarized for each post-Baseline assessment after Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
Millimoles per liter
  Chloride; Week 18; n=38, 34, 13, 12 | 1.9 (2.75) | 1 (2.5) | 1.8 (2.41) | 0.5 (2.94)
  Chloride; Week 24; n=35, 33, 12, 11 | 2 (2.33) | 0.7 (2.73) | 2.9 (2.81) | -0.2 (3.52)
  Chloride; Week 30; n=13, 10, 3, 2 | 1.9 (2.72) | 0.3 (2.87) | 5.3 (3.21) | 3 (0)
  Chloride; Week 36; n=10, 7, 2, 2 | 1.3 (2.11) | -0.1 (2.54) | 4.5 (6.36) | 1 (0)
  Chloride; Week 42; n=9, 6, 1, 2 | 1.3 (2.78) | 0 (2) | 10 (NA) — System value of NA indicates not applicable (too few participants). | 0.5 (0.71)
  Chloride; Week 48; n=6, 6, 0, 2 | 1.3 (2.34) | -1 (3.16) | NA (NA) — System value of NA indicates not applicable (too few participants). | 0 (0)
  Chloride; PT Week 4; n=33, 34, 11, 11 | 0.5 (2.69) | 0.2 (2.54) | 0.6 (2.29) | -1.5 (2.25)
  Bicarbonate; Week 18; n=38, 34, 13,12 | -0.3 (2.18) | -1 (2.16) | -1.2 (2.27) | 0 (2.95)
  Bicarbonate; Week 24; n=35, 33, 12,11 | -1 (2.41) | -1.2 (2.21) | -1.8 (2.41) | -0.4 (3.35)
  Bicarbonate; Week 30; n=13, 10, 3, 2 | 0.4 (2.33) | -2.2 (4.02) | -1.3 (1.53) | -2 (2.83)
  Bicarbonate; Week 36; n=10, 7, 2, 2 | -0.9 (2.92) | 0.1 (1.86) | -2.5 (2.12) | -1.5 (2.12)
  Bicarbonate; Week 42; n=9, 6, 1, 2 | -0.7 (1.73) | -0.2 (2.04) | -4 (NA) — System value of NA indicates not applicable (too few participants). | -1 (2.83)
  Bicarbonate; Week 48; n=6, 6, 0, 2 | -1 (1.67) | -1.3 (2.66) | NA (NA) — System value of NA indicates not applicable (too few participants). | -0.5 (3.54)
  Bicarbonate; PT Week 4; n=33, 34, 11,11 | -0.7 (2.1) | -0.5 (2.46) | -0.9 (2.43) | 1 (3.07)
  Glucose; Week 18; n=38, 34, 13, 12 | -0.28 (1.326) | -0.13 (1.188) | -0.06 (0.702) | -0.23 (2.134)
  Glucose; Week 24; n=35, 33, 12, 11 | -0.33 (1.552) | 0.27 (2.986) | -0.23 (0.672) | -0.22 (1.349)
  Glucose; Week 30; n=13, 10, 3, 2 | 0.03 (1.383) | -0.26 (0.587) | -0.13 (0.252) | 0.9 (0.707)
  Glucose; Week 36; n=10, 7, 2, 2 | -0.38 (0.758) | -0.37 (1.09) | -0.1 (0.99) | -0.7 (0.283)
  Glucose; Week 42; n=9, 6, 1, 2 | -0.28 (1.663) | -0.12 (0.794) | 0.4 (NA) — System value of NA indicates not applicable (too few participants). | -0.15 (0.919)
  Glucose; Week 48; n=6, 6, 0, 2 | 0.25 (1.358) | -0.3 (0.867) | NA (NA) — System value of NA indicates not applicable (too few participants). | 4.55 (4.596)
  Glucose; PT Week 4; n=33, 34, 11, 11 | 0.24 (3.122) | 0.18 (0.684) | -0.12 (0.735) | -0.07 (1.234)
  Potassium; Week 18; n=38, 34, 13, 12 | -0.19 (0.399) | -0.24 (0.376) | -0.41 (0.236) | -0.2 (0.424)
  Potassium; Week 24; n=35, 33, 12, 11 | -0.13 (0.452) | -0.12 (0.459) | -0.34 (0.403) | -0.32 (0.494)
  Potassium; Week 30; n=13, 10, 3, 2 | -0.03 (0.48) | -0.23 (0.377) | -0.1 (0.2) | -0.1 (0.424)
  Potassium; Week 36; n=10, 7, 2, 2 | 0.24 (0.599) | -0.1 (0.365) | 0.15 (0.071) | 0.2 (0.424)
  Potassium; Week 42; n=9, 6, 1, 2 | -0.1 (0.555) | -0.2 (0.415) | -0.1 (NA) — System value of NA indicates not applicable (too few participants). | 0.1 (0.566)
  Potassium; Week 48; n=6, 6, 0, 2 | 0.1 (0.566) | -0.3 (0.322) | NA (NA) — System value of NA indicates not applicable (too few participants). | 0.05 (0.495)
  Potassium; PT Week 4; n=33, 34, 11,11 | -0.16 (0.382) | -0.13 (0.398) | -0.25 (0.532) | -0.1 (0.316)
  Sodium; Week 18; n=38, 34, 13, 12 | 0.7 (2.04) | 0.1 (2.27) | 0.7 (2.32) | 0.4 (3.37)
  Sodium; Week 24; n=35, 33, 12, 11 | 0.4 (1.86) | -0.1 (2.61) | 1.5 (2.24) | 0.4 (3.53)
  Sodium; Week 30; n=13, 10, 3, 2 | 1.1 (3.25) | -1.4 (2.72) | 1.3 (1.53) | 0 (1.41)
  Sodium; Week 36; n=10, 7, 2, 2 | 0.4 (2.67) | -0.7 (1.98) | 2 (2.83) | -0.5 (0.71)
  Sodium; Week 42; n=9, 6, 1, 2 | 0.4 (2.07) | -0.5 (1.38) | 3 (NA) — System value of NA indicates not applicable (too few participants). | -1.5 (0.71)
  Sodium; Week 48; n=6, 6, 0, 2 | -0.2 (2.14) | -1.2 (2.79) | NA (NA) — System value of NA indicates not applicable (too few participants). | -2.5 (3.54)
  Sodium; PT Week 4; n=33, 34, 11, 11 | -0.1 (2.3) | 0.1 (2.45) | 1.1 (2.47) | -0.5 (2.7)
  Inorganic phosphorus; Week 18; n=38,34,13,12 | -0.161 (0.1971) | -0.13 (0.1928) | -0.092 (0.1537) | -0.111 (0.2648)
  Inorganic phosphorus; Week 24; n=35,33,12,11 | -0.139 (0.2268) | -0.13 (0.2354) | -0.119 (0.1991) | -0.107 (0.2205)
  Inorganic phosphorus; Week 30; n=13,10,3,2 | -0.156 (0.1644) | -0.118 (0.2071) | -0.267 (0.2023) | -0.225 (0.1768)
  Inorganic phosphorus; Week 36; n=10,7,2,2 | -0.121 (0.2564) | -0.167 (0.1906) | -0.195 (0.0495) | -0.125 (0.2475)
  Inorganic phosphorus; Week 42; n=9,6,1,2 | -0.08 (0.2248) | -0.108 (0.0794) | -0.15 (NA) — System value of NA indicates not applicable (too few participants). | -0.1 (0.3536)
  Inorganic phosphorus; Week 48; n=6,6,0,2 | -0.167 (0.1715) | -0.108 (0.1665) | NA (NA) — System value of NA indicates not applicable (too few participants). | -0.35 (0.0707)
  Inorganic phosphorus; PT Week 4;n=33,34,11,11 | -0.084 (0.2375) | -0.003 (0.2162) | 0.009 (0.0798) | -0.085 (0.2247)
  Urea/BUN; Week 18; n=38, 34, 13, 12 | -0.19 (1.166) | -0.23 (1.403) | -0.49 (1.233) | -0.25 (1.688)
  Urea/BUN; Week 24; n=35, 33, 12, 11 | -0.22 (1.263) | -0.55 (1.252) | -0.43 (1.106) | 0.02 (2.007)
  Urea/BUN; Week 30; n=13, 10, 3, 2 | 0.69 (1.107) | -0.16 (1.027) | -0.5 (1.082) | -0.5 (0)
  Urea/BUN; Week 36; n=10, 7, 2, 2 | 0.65 (1.775) | 0.04 (1.172) | -0.15 (0.636) | -0.25 (1.061)
  Urea/BUN; Week 42; n=9, 6, 1, 2 | 0.34 (1.65) | 0.5 (1.239) | 0.5 (NA) — System value of NA indicates not applicable (too few participants). | -0.5 (1.414)
  Urea/BUN; Week 48; n=6, 6, 0, 2 | 0.67 (1.353) | 0.4 (1.607) | NA (NA) — System value of NA indicates not applicable (too few participants). | -0.5 (0.707)
  Urea/BUN; PT Week 4; n=33, 34, 11,11 | 0.35 (1.284) | -0.19 (1.311) | -0.62 (1.012) | -0.47 (0.969)

39. Secondary Outcome: Mean Change From Baseline in Creatinine Clearance at the Indicated Time Points After Week 12
Description: Blood samples were collected for the measurement of estimated creatinine clearance by Cockcroft-Gault formula at the Baseline, Weeks 1, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, 48 and PT FU Weeks 4. Change from Baseline in the estimated creatinine clearance values are summarized for each post-Baseline assessment after Week 12. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Time Frame: Baseline (Week 0) and Weeks 18, 24, 30, 36, 42, 48 and PT FU Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Number analyzed (Participants) | 41 | 40 | 17 | 13
mL/min
  Creatinine clearance; Week 18; n=38, 34, 13, 12 | -0.1 (17.36) | -1.1 (20.69) | -2.5 (16.25) | -4.3 (19.37)
  Creatinine clearance; Week 24; n=35, 33, 12, 11 | -1.9 (16.77) | -1 (18.53) | -4.1 (15.11) | -6.1 (19.05)
  Creatinine clearance; Week 30; n=13,10,3,2 | -4.8 (13.91) | -10.4 (14.41) | -3.7 (13.58) | 7 (0)
  Creatinine clearance; Week 36; n=10,7,2,2 | -11 (23.3) | -8.1 (13.28) | -1 (29.7) | 1.5 (9.19)
  Creatinine clearance; Week 42; n=9, 6,1,2 | -6.1 (16.86) | -13.3 (16.13) | 9 (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | -1.5 (0.71)
  Creatinine clearance; Week 48; n=6, 6,0,2 | 3.2 (10.23) | -15.8 (16.18) | NA (NA) — The mean and standard deviation could not be determined (not reached) because too few participants experienced the event (system value of NA indicates not applicable for the mean and the standard deviation). | -4 (11.31)
  Creatinine clearance; PT Week 4; n=33,34,11,11 | -1.5 (34.53) | -1.3 (23.85) | -2.7 (11.38) | -5.3 (13.95)

40. Secondary Outcome: Correlation of Individual GSK2336805 Dose With Week 4 Plasma AUC(0-tau) Versus eRVR Status
Description: Correlation of individual GSK2336805 40 mg and 60 mg with Week 4 plasma AUC(0-tau) versus eRVR Status (eRVR and no eRVE) was performed. eRVR is defined as plasma HCV RNA <LLOQ and target not detected at Weeks 4 and 12. AUC (0-tau) is area under the concentration-time curve over the dosing interval. As defined in the RAP for this protocol, correlations between GSK2336805 dose, and selected pharmacokinetic parameters and virological outcomes was analyzed only with graphical presentations to facilitate clinical interpretation and data summarization. These data were also provided in by-participant data listings. Therefore, no statistical summary tables are available.
Time Frame: Week 4 and Week 12
Population: Intensive PK Population
Groups:
- GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV: Participants with chronic G1 and G4 HCV infection received GSK2336805 60 mg orally (30 mg x 2 tablets) once daily in the morning with food in combination with antiviral therapy (PEG+RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was 180 µg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken orally in 2 divided doses with food.
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV
Number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Correlation of Individual GSK2336805 Dose With Week 4 Plasma Cmax, Ctau, C0 Versus eRVR Status
Description: Correlation of Individual GSK2336805 40 mg and 60 mg dose with Week 4 maximum plasma concentration (Cmax), pre-dose concentration (C0), concentration at the end of the dosing interval (Ctau) versus eRVR status (eRVR and no eRVR) was performed. eRVR is defined as plasma HCV RNA <LLOQ and target not detected at Weeks 4 and 12. As defined in the RAP for this protocol, correlations between GSK2336805 dose, and selected PK parameters and virological outcomes was analyzed only with graphical presentations to facilitate clinical interpretation and data summarization. These data were also provided in by-participant data listings. Therefore, no statistical summary tables are available.
Time Frame: Week 4 and Week 12
Population: Intensive PK Population
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Correlation of Individual GSK2336805 Dose With Week 4 Plasma AUC(0-tau) Versus RVR Status
Description: Correlation of individual GSK2336805 40 mg and 60 mg with Week 4 plasma AUC(0-tau) versus eRVR Status (RVR and no eVE) was performed. RVR is defined as plasma HCV RNA <LLOQ and target not detected 4 weeks after initiation of therapy. AUC (0-tau) is area under the concentration-time curve over the dosing interval. As defined in the RAP for this protocol, correlations between GSK2336805 dose, and selected PK parameters and virological outcomes was analyzed only with graphical presentations to facilitate clinical interpretation and data summarization. These data were also provided in by-participant data listings. Therefore, no statistical summary tables are available.
Time Frame: Week 4
Population: Intensive PK Population
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Correlation of Individual GSK2336805 Dose With Week 4 Plasma Cmax, Ctau, C0 Versus RVR Status
Description: Correlation of Individual GSK2336805 40 mg and 60 mg dose with Week 4 maximum plasma concentration (Cmax), pre-dose concentration (C0), concentration at the end of the dosing interval (Ctau) versus RVR status (RVR and no RVR) was performed. RVR is defined as plasma HCV RNA <LLOQ and target not detected 4 weeks after initiation of therapy. As defined in the RAP for this protocol, correlations between GSK2336805 dose, and selected PK parameters and virological outcomes was analyzed only with graphical presentations to facilitate clinical interpretation and data summarization. These data were also provided in by-participant data listings. Therefore, no statistical summary tables are available.
Time Frame: Week 4
Population: Intensive PK Population
Groups:
- GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV: Participants with chronic G1 HCV infection received GSK2336805 60 mg orally (30 mg x 2 tablets) once daily in the morning with food in combination with antiviral therapy (PEG+RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was 180 µg once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken orally in 2 divided doses with food.
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: Correlation of Individual GSK2336805 Dose With Pre-dose Plasma Concentration at Week 4 and Week 12 Versus eRVR Status
Description: Correlation of individual GSK2336805 dose with pre-dose plasma concentration at Week 4 and Week 12 versus eRVR status was performed. eRVR is defined as plasma HCV RNA <LLOQ and target not detected at Weeks 4 and 12. The PK/Pharmacodynamic (PD) analysis population comprised of all participants with available PD measures (e.g., safety and/or efficacy data) and with evaluable GSK2336805 plasma concentration data considered suitable for investigation of relationship with the PD measures. As defined in the RAP for this protocol, correlations between GSK2336805 dose, and selected PK parameters and virological outcomes was analyzed only with graphical presentations to facilitate clinical interpretation and data summarization. These data were also provided in by-participant data listings. Therefore, no statistical summary tables are available.
Time Frame: Week 4 and Week 12
Population: PK/PD Analysis Population
Groups:
- GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV: Participants with chronic G1 HCV infection received GSK2336805 60 mg orally (30 mg x 2 tablets) once daily in the morning with food in combination with antiviral therapy (PEG+RIBA) for 12 weeks followed by PEG and RIBA alone for either 12 or 36 weeks based on eRVR achievement. PEG dose was 180 ug once weekly SC injection and the RIBA dose was 1000 mg orally (200 mg x 5 capsules) (if body weight was <75 kg) or 1200 mg orally (200 mg x 6 capsules) (if body weight was >=75 kg) taken orally in 2 divided doses with food.
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV
Number analyzed (Participants) | 0 | 0

45. Secondary Outcome: Correlation GSK2336805 Pre-dose Plasma Concentration on Day 2 Versus Reduction in HCV RNA on Day 2
Description: Correlation GSK2336805 pre-dose plasma concentration (ng/mL) on Day 2 versus reduction in HCV RNA (log IU/mL) on Day 2 was performed. As defined in the RAP for this protocol, correlations between GSK2336805 dose, and selected PK parameters and virological outcomes was analyzed only with graphical presentations to facilitate clinical interpretation and data summarization. These data were also provided in by-participant data listings. Therefore, no statistical summary tables are available.
Time Frame: Day 2
Population: PK/PD Analysis Population
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 and Genotype 4 HCV
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs and non-SAEs were collected from the start of study treatment until the follow-up contact (up to 20 study weeks).
Description: SAEs and non-SAEs were collected in participants of the safety population, comprised of all participants who had received at least one dose of study medication (GSK2336805 or telaprevir).
Arm/Group | GSK2336805 40 mg, Genotype 1 HCV | GSK2336805 60 mg, Genotype 1 HCV | Telaprevir, Genotype 1 HCV | GSK2336805 60 mg, Genotype 4 HCV
Serious Adverse Events (participants affected / at risk) | 2/41 | 2/40 | 3/17 | 1/13
Other Adverse Events (participants affected / at risk) | 41/41 | 38/40 | 17/17 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2336805 40 mg, Genotype 1 HCV (N=41) | GSK2336805 60 mg, Genotype 1 HCV (N=40) | Telaprevir, Genotype 1 HCV (N=17) | GSK2336805 60 mg, Genotype 4 HCV (N=13)
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Injection site abscess (Infections and infestations) | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2336805 40 mg, Genotype 1 HCV (N=41) | GSK2336805 60 mg, Genotype 1 HCV (N=40) | Telaprevir, Genotype 1 HCV (N=17) | GSK2336805 60 mg, Genotype 4 HCV (N=13)
Hypertension (Vascular disorders) | 3 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 5 | 1 | 0 | 1
Chills (General disorders) | 5 | 0 | 1 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 9 | 12 | 7 | 4
Feeling hot (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 8 | 9 | 3 | 8
Injection site bruising (General disorders) | 0 | 0 | 1 | 1
Injection site erythema (General disorders) | 6 | 3 | 1 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 1
Injection site pruritus (General disorders) | 0 | 2 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1
Injury associated with device (General disorders) | 0 | 0 | 0 | 1
Irritability (General disorders) | 4 | 0 | 0 | 2
Mucosal dryness (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 4 | 0 | 2 | 0
Pyrexia (General disorders) | 11 | 8 | 5 | 2
Temperature intolerance (General disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 5 | 3 | 1 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 4 | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 7 | 8 | 0 | 3
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 1 | 0 | 1
Nervousness (Psychiatric disorders) | 3 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Gingival injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0
International normalised ratio decreased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 2 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 22 | 14 | 9 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Eosinopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 6 | 10 | 6 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 5 | 2 | 0 | 1
Monocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 12 | 12 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 5 | 4 | 1
Disturbance in attention (Nervous system disorders) | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 5 | 2 | 1
Dysgeusia (Nervous system disorders) | 2 | 2 | 1 | 1
Headache (Nervous system disorders) | 15 | 14 | 5 | 4
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 2 | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 1 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 3 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 3
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 4 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 8 | 7 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 4 | 4 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4 | 3 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 5 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5 | 2 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 6 | 4 | 7 | 0
Rash (Skin and subcutaneous tissue disorders) | 8 | 5 | 7 | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 4 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 7 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 1 | 0
Body tinea (Infections and infestations) | 1 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.